## The GlaxoSmithKline group of companies

| Division | ŀ | Worldwide Development |
|--------------------|---|-----------------------------------|
| Information Type : | | Reporting and Analysis Plan (RAP) |

| Title | : | Reporting and Analysis Plan for Study 204958: An open-label, randomised, three arm, single dose, multi-centre, parallel group study in healthy subjects to compare the pharmacokinetics of subcutaneous mepolizumab when delivered as a liquid drug product in a safety syringe or an auto injector with a reconstituted lyophilised drug product from a vial. |
|---|---|---|
| <b>Compound Number</b> | : | SB-240563 |
| Effective Date | : | 03-AUG-2017 |

## **Description:**

- The purpose of this RAP is to describe the planned statistical analyses and associated data displays to be included in the Clinical Study Report for Protocol 204958.
- This RAP defines the content of the final Statistical Analysis Complete (SAC) deliverable.

#### **Author's Name and Functional Area:**

| PPD | 19-JUL-2017 |
|------------------------------|-------------|
| Manager, Clinical Statistics | 19-JUL-2017 |

## Reviewed/Agreed by:

| PPD [1] | Director, Clinical Pharmacology | 19-JUL-2017 |
|---------|------------------------------------------|-------------|
| PPD [2] | Product Physician Lead | 18-JUL-2017 |
| PPD [1] | Clinical Operations | 21-JUL-2017 |
| PPD [1] | Clinical Investigational Lead | 03-AUG-2017 |
| PPD [1] | Director, CMO GCSP SERM | 02-AUG-2017 |
| PPD [1] | Data Quality Lead | 19-JUL-2017 |
| PPD [1] | Programmer/Analyst, Clinical Programming | 20-JUL-2017 |
| PPD [1] | Manager, Clinical Programming | 19-JUL-2017 |

## Final Technical Approval by:

| PPD [1] | 02 AUC 2017 |
|-------------------------------|-------------|
| Director, Clinical Statistics | 03-AUG-2017 |

<sup>[1]</sup> Approval captured electronically within the C.A.R.S system.

Copyright 2017 the GlaxoSmithKline group of companies. All rights reserved. Unauthorised copying or use of this information is prohibited.

<sup>[2]</sup> Approval via email.

## **TABLE OF CONTENTS**

| | | | PAGE |
|---|---|---|---|
| 1. | REPO | RTING & ANALYSIS PLAN SYNPOSIS | 4 |
| 2. | SUMM<br>2.1.<br>2.2.<br>2.3.<br>2.4. | IARY OF KEY PROTOCOL INFORMATION Changes to the Protocol Defined Statistical Analysis Plan Study Objective(s) and Endpoint(s). Study Design Statistical Hypotheses. | 6<br>6 |
| 3. | PLANN<br>3.1.<br>3.2. | NED ANALYSESInterim AnalysesFinal Analyses | 8 |
| 4. | ANALY<br>4.1. | YSIS POPULATIONSProtocol Deviations | |
| 5. | | IDERATIONS FOR DATA ANALYSES AND DATA HANDLING | 11 |
| 6. | STUD'<br>6.1. | Y POPULATION ANALYSES | |
| 7. | PHARI<br>7.1.<br>7.2.<br>7.3.<br>7.4. | MACOKINETIC ANALYSES Overview of Planned Pharmacokinetic Analyses Drug Concentration Measures Derived Plasma Pharmacokinetic Parameters Planned Primary Pharmacokinetic Analyses | 12<br>13 |
| 8. | SAFE1<br>8.1.<br>8.2. | TY ANALYSIS Overview of Planned Adverse Event Analyses | 16<br>17 |
| 9. | IMMUN<br>9.1. | NOGENICITY<br>Overview of Planned Immunogenicity Analyses | |
| 10. | 10.1. | DRATORY STATISTICAL ANALYSES | 20<br>20<br>20 |
| 11. | REFE | RENCES | <mark>22</mark> |
| 12. | APPEN<br>12.1.<br>12.2. | Appendix 1: Time & Events | 24<br>24<br>28 |

## CONFIDENTIAL

| 12.3. | Appendix | x 3: Data Display Standards & Handling Conventions | 29 |
|---|---|---|---|
| | 12.3.1. | | |
| | 12.3.2. | Baseline Definition & Derivations | |
| | | 12.3.2.1. Baseline Definitions | |
| | | 12.3.2.2. Derivations and Handling of Missing Baseline | |
| | | Data | 30 |
| | 12.3.3. | Reporting Process & Standards | |
| 12.4. | | x 4: Derived and Transformed Data | |
| | 12.4.1. | General | |
| | 12.4.2. | Study Population | |
| | 12.4.3. | Pharmacokinetics | |
| | 12.4.4. | Safety | |
| | 12.4.5. | | |
| 12.5. | Appendix | x 5: Premature Withdrawals & Handling of Missing Data | |
| | 12.5.1. | | |
| | 12.5.2. | Handling of Missing Data | 35 |
| | | 12.5.2.1. Handling of Missing and Partial Dates | |
| 12.6. | Appendix | x 6: Values of Potential Clinical Importance | |
| | 12.6.1. | · | |
| 12.7. | Appendix | x 7: Multicenter Studies | <mark>38</mark> |
| 12.8. | | x 8: Examination of Covariates, Subgroups & Other Strata | |
| | 12.8.1. | Handling of Covariates | 39 |
| | 12.8.2. | Handling of Subgroups | 39 |
| 12.9. | Appendix | x 9: Abbreviations & Trade Marks | 40 |
| | 12.9.1. | | |
| | 12.9.2. | Trademarks | |
| 12.10. | | x 10: List of Data Displays | |
| | | Study Population Tables | |
| | | Pharmacokinetic Figures | |
| | | Pharmacokinetic Tables | |
| | | Safety Tables | |
| | | Immunogenicity Tables | |
| | | Exploratory Figures | |
| | | Exploratory Tables | |
| | | ICH and Other Listings | |
| 12.11. | Appendix | x 11: Example Mock Shells for Data Displays | 60 |

# 1. REPORTING & ANALYSIS PLAN SYNPOSIS

| Overview | Key Elements of the Reporting and Analysis Plan (RAP) |
|---|---|
| Purpose | This RAP defines the content of the final Statistical Analysis Complete (SAC) deliverable. |
| Protocol | <ul> <li>This RAP is based on protocol amendment 2 dated 17-NOV-2016<br/>[GlaxoSmithKline Document Number: 2016N275057_02].</li> </ul> |
| Primary Objective / Endpoint | To compare the pharmacokinetics of subcutaneous mepolizumab following a single dose of the liquid drug product in safety syringe with the lyophilized drug product. |
| | <ul> <li>Mepolizumab PK parameters: Cmax, AUC(0-t) and AUC(0-∞)</li> </ul> |
| | <ul> <li>To compare the pharmacokinetics of subcutaneous mepolizumab following a<br/>single dose of the liquid drug product in autoinjector with the lyophilized drug<br/>product.</li> </ul> |
| | <ul> <li>Mepolizumab PK parameters: Cmax, AUC(0-t) and AUC(0-∞)</li> </ul> |
| Study<br>Design | Single dose, randomised, open-label, multi-centre, parallel group study in healthy subjects. |
| | Two test drug products (mepolizumab liquid drug product in an autoinjector and mepolizumab liquid drug product in a safety syringe) will be compared with a reference drug product (reconstituted lyophilised mepolizumab drug product from a vial). |
| | Approximately 243 healthy subjects will be randomised to obtain at least 216 completed subjects. |
| | <ul> <li>Mepolizumab injection site (upper arm, abdomen or thigh) and treatment will be<br/>assigned randomly. The randomisation will be stratified by body weight (&lt;70kg,<br/>70-&lt;80kg and ≥80kg).</li> </ul> |
| | Subjects will be followed for 85 days following drug administration. |
| Analysis<br>Population | Primary: Pharmacokinetic Population. Comprise all subjects receiving study drug for whom a pharmacokinetic sample was obtained and analysed. |
| Hypothesis | <ul> <li>No formal hypothesis will be tested. For AUC(0-t), AUC(0-∞) and Cmax, point estimates and corresponding two-sided 90% confidence intervals will be constructed for the ratio of the geometric mean of each test treatment to the geometric mean of the reference treatment, µ(test)/µ(reference).</li> </ul> |
| Primary<br>Analyses | • The analysis for each treatment comparison will be conducted excluding subjects receiving the test treatment that is not relevant for that comparison. The parameters AUC(0-t), AUC(0-∞) and Cmax will be loge transformed and analysed separately using a fixed effects model, including treatment group and injection site (upper arm, abdomen, thigh) as categorical variables and baseline weight as a continuous covariate fitted on the loge scale. Point estimates and associated two-sided 90% CIs will be constructed for the differences between the test and reference treatments on the loge scale; these will be backtransformed to provide point estimates and two-sided 90% CIs for the ratio of each of the test treatments to the reference treatment on the original scale. |

## CONFIDENTIAL

| Overview | Key Elements of the Reporting and Analysis Plan (RAP) |
|---|---|
| Secondary Analyses Safety data will be presented in tabular and/or graphical format and summ descriptively according to GSK's Integrated Data Standards Library (IDSL) standards. | |
| Exploratory<br>Analyses | <ul> <li>Ratio to baseline blood eosinophils will be log transformed and compared<br/>between treatments at each visit using a mixed model repeated measures<br/>analysis, adjusting for the covariates of baseline blood eosinophil count (log<br/>scale) and baseline weight (log scale). Visit and injection site (upper arm,<br/>abdomen, thigh) will be fitted as categorical variables with the effect of treatment<br/>group and baseline blood eosinophil count varying at each visit (i.e.<br/>visit-by-baseline and visit-by-treatment interactions will be included in the<br/>model).</li> </ul> |

## 2. SUMMARY OF KEY PROTOCOL INFORMATION

## 2.1. Changes to the Protocol Defined Statistical Analysis Plan

Three additional analysis populations were defined for reporting screen failures, inclusion exclusion criteria deviations and blood eosinophils. These are described in Section 4.

There are no other changes to the protocol defined statistical analysis plan.

# 2.2. Study Objective(s) and Endpoint(s)

| Ob | jectives | Endpoints | |
|---|---|---|---|
| Pri | mary Objectives | Pri | imary Endpoints |
| • | To compare the pharmacokinetics of subcutaneous mepolizumab following a single dose of the liquid drug product in safety syringe with the lyophilized drug product. | • | Mepolizumab PK parameters:<br>Cmax, AUC(0-t) and AUC(0-∞) |
| • | To compare the pharmacokinetics of subcutaneous mepolizumab following a single dose of the liquid drug product in autoinjector with the lyophilized drug product. | • | Mepolizumab PK parameters:<br>Cmax, AUC(0-t) and AUC(0-∞) |
| Se | condary Objectives | Se | condary Endpoints |
| • | To assess additional pharmacokinetic parameters following mepolizumab subcutaneous administration of the liquid drug product in autoinjector or the liquid drug product in safety syringe in comparison with the lyophilized drug product, as data permit. | • | Mepolizumab PK parameters: tmax, CL/F, Vd/F, λz, t ½, tlast, %AUCex |
| • | To assess the safety and tolerability of mepolizumab following a single SC dose of the liquid drug product in autoinjector or the liquid drug product in safety syringe in comparison with the lyophilised drug product. | • | Adverse events (AEs), serious adverse events (SAEs), including systemic reactions and injection site reactions Haematology and Clinical Chemistry Vital signs 12-lead ECG |
| • | To assess the immunogenicity of mepolizumab following a single SC dose of the liquid drug product in autoinjector or the liquid drug product in safety syringe in | • | Frequency of positive anti-mepolizumab binding antibodies and neutralizing antibodies |

| Objectives | Endpoints |
|---|---|
| comparison with the lyophilised drug product. | |
| Exploratory Objectives | Exploratory Endpoints |
| To evaluate mepolizumab pharmacodynamic effects on blood eosinophil count following a single SC dose of the liquid drug product in safety syringe or the liquid drug product in autoinjector in comparison with the lyophilised drug product. | Ratio to baseline in blood eosinophil count over time |
| To evaluate safety syringe and autoinjector use & functionality. | User and device errors |

## 2.3. Study Design



| Overview of S | Overview of Study Design and Key Features |
|---|---|
| Treatment Assignment | |
| | Mepolizumab injection site and treatment will be assigned randomly and the randomization schedule will be generated using GSK validated randomisation software RandAll NG. Allocations to injection site and treatment will be made centrally via an interactive response system (IRS). |
| <ul> <li>The randomisation will be stratified by body weight (&lt;70kg, 70-&lt;80kg and ≥80kg) measured on Day -1. Subjects will be randomised in a 1:1:1 ratio to one of 3 different injection sites (upper arm, abdomen and thigh) and in a ratio to one of 3 mepolizumab treatments (liquid drug product in an autoinjector, liquid drug product in a safety syringe and reconstituted lyophilised drug product from a vial). A minimum of 27 subjects will be randomised within each of the 3 body weight strata to ensure at least 3 subjects within each body weight strata, injection site and mepolizumab treatment combination.</li> </ul> | |
| Time and events | See Appendix 1: Time & Events. |
| Interim<br>Analysis | No interim analyses are planned. |

## 2.4. Statistical Hypotheses

This study is designed to evaluate mepolizumab PK comparability following a single SC administration, i.e. the relative bioavailability, between

- The liquid drug product from the autoinjector (test) and the reconstituted lyophilised drug product from the vial (reference)
- The liquid drug product from the safety syringe (test) and the reconstituted lyophilised drug product from the vial (reference)

For AUC(0-t), AUC(0- $\infty$ ) and Cmax, point estimates and corresponding two-sided 90% confidence intervals will be constructed for the ratio of the geometric mean of each test treatment to the geometric mean of the reference treatment,  $\mu(\text{test})/\mu(\text{reference})$ . No formal hypothesis will be tested. However, interpretation of the comparability of the autoinjector and safety syringe with the reconstituted lyophilised drug product will be guided by a two-sided 90% confidence interval (CI) for  $\mu(\text{test})/\mu(\text{reference})$  in the range (0.80, 1.25) for AUC(0-t), AUC(0- $\infty$ ) and Cmax.

## 3. PLANNED ANALYSES

## 3.1. Interim Analyses

No interim analyses are planned.

## 3.2. Final Analyses

The final planned analyses will be performed after the completion of the following steps:

- 1. All subjects have completed the study as defined in the protocol.
- 2. All required database cleaning activities have been completed and final database release and database freeze (DBF) has been declared by Data Management.
- 3. A review has taken place to identify any subjects with a discrepancy between randomised treatment and actual treatment received. This information will be included in the SDTM datasets at database freeze (DBF).
- 4. Treatment allocations have been unblinded via the RandAll NG system, as described in SOP\_54840. Although the study is open-label, treatment allocations remain blinded in the RandAll NG system until source data lock (SDL) as per SOP\_54840.

## 4. ANALYSIS POPULATIONS

| Population | Definition / Criteria | Analyses Evaluated |
|---|---|---|
| All Subjects<br>Enrolled | Comprise all subjects enrolled and for whom a record exists in the data base. | Screen failures |
| Randomised | Comprise all randomised subjects | Listing of exclusions<br>from study<br>populations |
| All Treated<br>Subjects (Safety) | <ul> <li>Comprise all subjects who receive mepolizumab.</li> <li>This population will be based on the treatment the subject actually received.</li> </ul> | <ul><li>Study population</li><li>Safety</li><li>Immunogenicity</li><li>User/device errors</li></ul> |
| Pharmacokinetic<br>(PK) | <ul> <li>Subjects in the 'All Treated Subjects' population for whom a PK sample was obtained and analysed.</li> <li>This population will be based on the treatment the subject actually received.</li> </ul> | PK, including primary analysis |
| Pharmacodynamic (PD) | <ul> <li>Subjects in the 'All Treated Subjects' population who had a baseline PD measurement and at least one post-treatment PD measurement.</li> <li>This population will be based on the treatment the subject actually received.</li> </ul> | Blood eosinophils |

#### NOTES:

 Please refer to Appendix 10: List of Data Displays which details the population to be used for each displays being generated.

#### 4.1. Protocol Deviations

- Protocol deviations will be tracked by the study team throughout the conduct of the study in accordance with the Protocol Deviation Management Plan.
  - o Data will be reviewed prior to DBF to ensure all important deviations are captured and categorised on the protocol deviations dataset.
  - This dataset will be the basis for the summaries and listings of protocol deviations.
- Important protocol deviations (including deviations related to study inclusion/exclusion criteria, conduct of the trial, subject management or subject assessment) will be summarised and listed.
- A separate summary and listing of all inclusion/exclusion criteria deviations will also be provided. This summary will be based on data as recorded on the inclusion/exclusion page of the eCRF.

# 5. CONSIDERATIONS FOR DATA ANALYSES AND DATA HANDLING CONVENTIONS

Table 1 provides an overview of appendices within the RAP for outlining general considerations for data analyses and data handling conventions.

Table 1 Overview of Appendices

| Section | Component |
|---|---|
| Section 12.1 | Appendix 1: Time & Events |
| Section 12.2 | Appendix 2: Treatment States and Phases |
| Section 12.3 | Appendix 3: Data Display Standards & Handling Conventions |
| | Study Treatment & Injection Site Descriptors |
| | Baseline Definition & Derivations |
| | Reporting Process & Standards |
| Section 12.4 | Appendix 4: Derived and Transformed Data |
| | General |
| | Study Population |
| | Pharmacokinetics |
| | Safety |
| | Blood Eosinophils |
| Section 12.5 | Appendix 5: Premature Withdrawals & Handling of Missing Data |
| Section 12.6 | Appendix 6: Values of Potential Clinical Importance |
| Section 12.7 | Appendix 7: Multicenter Studies |
| Section 12.8 | Appendix 8: Examination of Covariates, Subgroups & Other Strata |
| Section 12.9 | Appendix 9: Abbreviations & Trade Marks |
| Section 12.10 | Appendix 10: List of Data Displays |

## 6. STUDY POPULATION ANALYSES

## 6.1. Overview of Planned Analyses

The study population analyses will be based on the "All Treated Subjects (Safety)" population.

Table 2 provides an overview of the planned study population analyses. Full details of the data displays to be presented are given in Appendix 10: List of Data Displays.

Table 2 Overview of Planned Study Population Analyses

| Display Type | Data | Displays Gene | erated |
|---|---|---|---|
| | Table | Figure | Listing |
| Study Populations | Y | | Υ |
| Screen Failures | Y | | Υ |
| Randomisation | | | Υ |
| Subject Disposition | Y | | Υ |
| Important Protocol Deviations | Y | | Υ |
| Inclusion/Exclusion Criteria Deviations | | | Υ |
| Exposure to Study Treatment | | | Υ |
| Demographics | Y | | Υ |
| Past and Current Medical Conditions | Y | | Y |
| Family History of Cardiovascular Risk Factors | Y | | Y |
| Other Family History | | | Y |
| Smoking History | Y | | |
| Concomitant Medications | | | Y |

#### NOTES:

• Y = Yes display generated.

## 7. PHARMACOKINETIC ANALYSES

The primary objective of this study is to evaluate the PK comparability of the liquid drug product administered by both the autoinjector and safety syringe with the lyophilised drug product when reconstituted from the vial.

## 7.1. Overview of Planned Pharmacokinetic Analyses

The pharmacokinetic (PK) analyses will be based on the "Pharmacokinetic" population.

The planned primary statistical analysis is detailed in Section 7.4. Summaries of the PK concentration-time data and PK parameters are detailed in Section 7.2 and Section 7.3 respectively.

Table 3 provides an overview of the planned pharmacokinetic data displays. Full details of the data displays to be presented are given in Appendix 10: List of Data Displays.

Table 3 Overview of Planned Pharmacokinetic Analyses

| Endpoints | | | Un | transfor | med | | Log-Transformed | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Stats Analysis | | | Summ | ary | Indiv | idual | Stats | Analy | sis ( | Sum | mary | Individual | |
| | F | Т | L | F | Т | F | L | F | Т | L | F | Т | F | L |
| PK Plasma<br>Concentrations | | | | <b>Y</b> [1] [2] | Υ | Y [1] | Y | | | | | | | |
| Derived Plasma PK<br>Parameters | | | | | Υ | | Y | <b>Y</b> [3] | <b>Y</b> [3] | | <b>Y</b> [3] | Υ | | |

#### NOTES:

- T = Table, F = Figures, L = Listings, Y = Yes display generated.
- Stats Analysis = Represents TFL related to any formal statistical analyses (i.e. modelling) conducted.
- Summary = Represents TFL related to any summaries (descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data.
- 1. Linear and Semi-Log plots will be created on the same display.
- 2. Separate Mean (± SD) and Median plots will be generated.
- Cmax, AUC(0-t) and AUC(0-∞) only.

## 7.2. Drug Concentration Measures

Blood sampling time will be related to the start of dosing. Linear and semi-logarithmic individual plasma concentration-time profiles and mean (±SD) and median profiles will be plotted for each treatment.

Plasma concentrations of mepolizumab will be listed and summarised by treatment group and nominal time. Summaries, including mean (±SD) and median profile plots, will also be produced by treatment group and injection site, treatment group and baseline body weight category (<70kg, 70-<80kg and ≥80kg), and treatment group, injection site and baseline body weight category. Any subjects randomised in error to the incorrect weight strata will be summarised according to the stratum corresponding to their actual body weight. No formal statistical analysis of the body weight subgroups is planned.

Refer to Appendix 3: Data Display Standards & Handling Conventions, Section 12.3.3 Reporting Process & Standards.

#### 7.3. Derived Plasma Pharmacokinetic Parameters

- Mepolizumab pharmacokinetic parameters will be calculated by standard noncompartmental analysis according to current working practices (GUI\_51487 (4.0)) and using Phoenix.
- Calculations will be based on the actual sampling times recorded during the study.
- From the plasma concentration-time data, the pharmacokinetic parameters in Table 4
  will be determined for mepolizumab, as data permit, for each treatment and for each
  subject.

- Individual and geometric mean (95% CI) Cmax, AUC(0-t) and AUC(0-∞) will be plotted by treatment group, by treatment group and injection site, by treatment group and baseline body weight category (<70kg, 70-<80kg and ≥80kg), and by treatment group, injection site and baseline body weight category.
- All pharmacokinetic parameters will be listed and summarized descriptively by treatment group, by treatment group and injection site, by treatment group and baseline body weight category (<70kg, 70-<80kg and ≥80kg), and by treatment group, injection site and baseline body weight category.
- Any subjects randomised in error to the incorrect weight strata will be summarised
  according to the stratum corresponding to their actual body weight. No formal
  statistical analysis of the body weight subgroups is planned.
- Refer to Appendix 3: Data Display Standards & Handling Conventions, Section 12.3.3 Reporting Process & Standards.

Table 4 Derived Pharmacokinetic Parameters

| Parameter | Parameter Description |
|---|---|
| Cmax | Maximum observed plasma concentration |
| tmax | Time to Cmax |
| AUC(0-∞) | Area under the plasma concentration-time curve from time zero extrapolated to infinite time. |
| AUC(0-t) | Area under the plasma concentration-time curve from time zero to the time of the last quantifiable concentration. |
| AUC(0-week4) | Area under the plasma concentration-time from time zero to Week 4. |
| %AUCextrapolated | Percentage of AUC(0-∞) obtained by extrapolation |
| tlast | Last time point where the concentration is above the limit of quantification |
| CL/F | Apparent clearance |
| Vd/F | Apparent volume of distribution |
| λz | Terminal phase elimination rate constant. |
| | The number of points used to determine λz will also be reported. |
| t½ | Terminal phase half-life |

**NOTES:** Additional parameters may be included as required.

## 7.4. Planned Primary Pharmacokinetic Analyses

#### **Primary Statistical Analyses**

## Endpoint(s)

• Cmax, AUC(0-t), AUC(0-∞)

#### **Endpoint Derivation**

 Derivation of pharmacokinetic parameters will be according to current working practices (GUI\_51487 (4.0)).

#### **Handling of Missing Data**

 Analysis will be performed on all available data and no imputation will be performed for missing data.

## **Model Specification**

- Each test treatment (liquid formulation from the autoinjector or safety syringe) will be compared to the reference (reconstituted lyophilised powder from the vial).
- Separate models will be used for each treatment comparison, including only data from the
  relevant test treatment and the reference treatment. Data from the test treatment that is not
  relevant for that comparison will be excluded.
- The parameters Cmax, AUC(0-t), AUC(0-∞) will be loge transformed and analysed separately
  using a fixed effects analysis of covariance model, including treatment group and injection site
  (upper arm, abdomen, thigh) as categorical variables and baseline body weight as a
  continuous covariate fitted on the loge scale.
- The MIXED procedure in SAS will be used with the following options:-
  - The Kenward and Roger method for approximating the denominator degrees of freedom to correct for bias in the estimated variance-covariance.
  - The OBSMARGIN option on the LSMEANS statement in order to compute the adjusted geometric means with weights proportional to the input data set.

#### **Multiple Comparisons and Multiplicity**

 Each treatment comparison will be considered separately and no adjustment for multiplicity will be made.

#### Model Checking & Diagnostics

Distributional assumptions underlying the models used for analysis will be examined by
obtaining box plots and normal probability plots of the studentized residuals and plots of the
residuals versus the fitted values (i.e. checking the normality assumption and constant
variance assumption of the model respectively) to gain confidence that the model assumptions
are reasonable.

#### **Model Results Presentation**

For each PK parameter:-

- Adjusted geometric mean for each treatment group and standard error (loge scale).
- Point estimates and associated two-sided 90% confidence intervals for the ratio of each of the
  test treatments to the reference treatment (obtained by back-transforming estimates and 90%
  Cls for the treatment differences from the statistical model on the loge scale).

## 8. SAFETY ANALYSIS

The safety displays to be created as part of this RAP include all the required and relevant displays identified as per the IDSL Core Safety Statistical Displays.

Analysis of safety data will be based on the 'All Treated (Safety)" population.

All safety data will be presented using the treatment group descriptors defined in Section 12.3. In addition, a "Total Liquid" column will present the combined results from the liquid autoinjector and liquid safety syringe, and a "Total" column will present the combined results across all 3 randomised treatment groups.

## 8.1. Overview of Planned Adverse Event Analyses

Table 5 provides an overview of the planned analyses of adverse event data. Full details of the data displays to be presented are given in Appendix 10: List of Data Displays.

Table 5 Overview of Planned Adverse Event Analyses

| Endpoint / Parameter/ Display Type | | Absol | ute |
|---|---|---|---|
| | Sun | nmary | Individual |
| | Т | F | L |
| Adverse Events (AEs) | | | |
| All AEs by SOC | Υ | | Y |
| Common AEs by Overall Frequency <sup>[1]</sup> | Υ | | |
| No. of Subjects & No. of Occurrences of Common AEs by SOC and PT[1] | Υ | | |
| All AEs by SOC and Maximum Intensity | Υ | | |
| All Drug-Related AEs by SOC | Υ | | |
| All Drug-Related AEs by SOC and Maximum Intensity | Y | | |
| AEs by Highest Post Baseline Binding Antibody Result (see Section 9.1) | Y | | |
| AEs Leading to Withdrawal from Study by Overall Frequency | Υ | | Υ |
| AEs reported on the Day of Dosing[2] | Y | | Υ |
| Subject Numbers for Individual AEs | | | Υ |
| Relationship Between AE SOCs, PT & Verbatim Text | | | Υ |
| Serious and Other Significant AEs | | | |
| Fatal Serious AEs by Overall Frequency | Υ | | Υ |
| All Serious AEs by SOC | Y | | |
| Non-Fatal Serious AEs | | | Υ |
| Reasons for Considering as a Serious AE | | | Υ |
| Drug-Related Fatal Serious AEs by Overall Frequency | Υ | | |
| Drug-Related Serious AEs by SOC | Y | | |
| No. of Subjects & No. of Occurrences of All Serious AEs | Υ | | |
| Adverse Events of Special Interest (AESI) | | | |
| Anaphylaxis | Y | | Υ |
| Systemic Reactions – Allergic (Type I Hypersensitivity) and Other Systemic | Υ | | Y |
| Systemic Reactions – Allergic (Type I Hypersensitivity) | Y | | Υ |
| Systemic Reactions – Other Systemic | Y | | Υ |

| Endpoint / Parameter/ Display Type | | Absolute | |
|---|---|---|---|
| | Sun | nmary | Individual |
| | Т | F | L |
| Local Injection Site Reactions | Υ | | Υ |
| Opportunistic Infections | Υ | | Υ |
| Malignancies | Υ | | Y |
| Serious Cardiac, Vascular and Thromboembolic Events | Υ | | Υ |
| Serious Ischemic Events | Υ | | Y |

#### NOTES:

- T = Table, F = Figure, L = Listing, Y = Yes display generated, SOC = System Organ Class, PT = Preferred Term.
- Summary = Represents TFL related to any summaries (i.e. descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data.
- [1] Common AEs will be defined as AEs with frequency ≥3% (prior to rounding to nearest percent) in either the Total Liquid or Lyophilised Vial treatment groups.
- [2] AEs reported on the day of dosing will be defined as adverse events with a start date equal to the date of dosing.

## 8.1.1. Adverse Events of Special Interest

Adverse events of special interest (AESIs) are adverse events associated with the identified and potential risks of mepolizumab. AESIs reported by the investigator as anaphylaxis reactions, systemic reactions (further categorised by the investigator as either allergic (type I hypersensitivity) or other systemic reactions) and local injection site reactions are collected via targeted eCRF within the study.

AESIs of opportunistic infections, malignancies, serious cardiac vascular and thromboembolic (CVT) events and serious ischemic events will be identified from a list of relevant preferred terms maintained within a project level reference dataset created based on the MedDRA dictionary available at the time of database freeze for this study. Further details of how relevant preferred terms are identified are given in the Program Safety Analysis Plan (PSAP).

Separate summary tables showing the number and percent of subjects with each type of AESI, broken down by preferred term will be created.

For each type of AESI a profile summary table will be produced containing information including, but not be limited to, the number of occurrences of the event, event characteristics, time to onset, intensity, outcome and action taken.

Separate listings of AESIs identified by the investigator as anaphylaxis, allergic (type I hypersensitivity), other systemic reactions and local injection site reactions will be produced, as well as listings of opportunistic infections, malignancies, serious CVT events and serious ischemic events

# 8.2. Overview of Other Safety Analyses

Table 6 provides an overview of the planned analyses for laboratory data, ECG and vital signs. Full details of the data displays to be presented are given in Appendix 10: List of Data Displays.

Table 6 Overview of Other Safety Analyses

| Endpoint / Parameter/ Display Type | | Abs | olute | Change from BL | | |
|---|---|---|---|---|---|---|
| | Sum | mary | Individual | Sumr | nary | Individual |
| | Т | F | L | Т | F | L |
| Haematology | | | | | | |
| Haematology Changes from Baseline | | | | Υ | | |
| Haematology Shifts from Baseline Relative to Normal Range | | | | Y | | |
| Haematology Shifts from Baseline Relative to PCI Range | | | | Υ | | |
| Haematology Data for Subjects with Any Value of Potential Clinical Concern | | | Y | | | |
| Chemistry | | | | | | |
| Chemistry Changes from Baseline | | | | Υ | | |
| Chemistry Shifts from Baseline Relative to Normal Range | | | | Υ | | |
| Chemistry Shifts from Baseline Relative to PCI Range | | | | Υ | | |
| Chemistry Data for Subjects with Any Value of Potential Clinical Concern | | | Y | | | |
| ECG | | | | | | |
| ECG Findings | Υ | | | | | |
| Vital Signs | | | | | | |
| Vital Signs Change from Baseline | | | | Υ | | |

#### NOTES:

- T = Table, F = Figures, L = Listings, Y = Yes display generated. PCI = Potential Clinical Importance see Section 12.6
- Summary = Represents TFL related to any summaries (i.e. descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data.

#### 9. IMMUNOGENICITY

## 9.1. Overview of Planned Immunogenicity Analyses

For the immunogenicity assessment, two types of anti-drug antibody (ADA) assays will be performed, a binding anti-drug antibody assay and a neutralizing antibody assay.

For the binding assay, there will be a three tiered analysis: screening, confirmation and titration. The screening assay produces a result of positive or negative relative to a screening cut point. Positive samples continue with the confirmation assay, which also produces a result of positive or negative relative to a confirmation cut point. For positive confirmation samples, a titre value will also be obtained to quantify the degree of binding in a titration assay and the sample will be tested with the neutralizing assay, which also reports results as positive or negative.

The binding ADA results at each visit will be categorised as negative, transient positive (defined as a single confirmatory positive immunogenic response that does not occur at

the final study assessment) or persistent positive (defined as a confirmatory positive immunogenic response for at least 2 consecutive assessments excluding the screening visit, or a single result at the final study assessment). In addition, the highest post-baseline binding ADA confirmatory result obtained for a subject will be summarised. Subjects with both positive and negative results will be identified in the positive category. Summary statistics for the highest titre result will also be presented.

A summary of adverse events by highest post-baseline binding antibody result (as defined above) will be produced.

A summary of treatment emergent positive confirmatory binding ADA assays in the subset of subjects who did not have a positive confirmatory binding ADA assay prior to the dosing of study treatment will also be presented.

Neutralizing antibody assay results will be summarised by visit. In addition, the highest post-baseline neutralising assay result during the treatment period of the study will be summarised, with subjects with both positive and negative results identified in the positive category.

Immunogenicity data will be listed for subjects with at least one positive screening binding assay.

## 10. EXPLORATORY STATISTICAL ANALYSES

## 10.1. Blood Eosinophils

## 10.1.1. Overview of Planned Analyses for Blood Eosinophils

Blood eosinophil analyses will be based on the "Pharmacodynamic" population.

Blood eosinophil values will be log<sub>e</sub>-transformed prior to summary and analysis. Non-detectable values of 0 GI/L, will be replaced by half of the lowest observed detectable (non-zero) value in the study data set, prior to log transformation.

Table 7 provides an overview of the planned analyses for blood eosinophils. Full details of data displays to be presented are given in Appendix 10: List of Data Displays.

Table 7 Overview of Planned Analyses for Blood Eosinophils

| Endpoint | | | Un | transfo | med | | Log-Transformed | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Stat | Stats Analysis | | Summ | ary | Indiv | idual | Stats | Analy | sis | Sum | mary | Individual | |
| | F | Т | L | F | Т | F | F L | | T L | | F | Т | F | L |
| Absolute Blood<br>Eosinophils | | | | | Υ | | | | | | | Υ | | |
| Ratio to Baseline<br>Blood Eosinophils | | | | | Υ | | | Y | Y | | | Υ | | |

#### NOTES:

- T = Table, F = Figures, L = Listings, Y = Yes display generated.
- Stats Analysis = Represents TFL related to any formal statistical analyses (i.e. modelling) conducted.
- Summary = Represents TFL related to any summaries (descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data.

#### 10.1.2. Planned Analysis of Blood Eosinophils

#### **Blood Eosinophil Analyses**

#### Endpoint(s)

Ratio to Baseline Blood Eosinophils

#### **Model Specification**

- Ratio to Baseline Blood Eosinophils will be loge transformed and compared between treatments using a mixed model repeated measures analysis, adjusting for baseline blood eosinophil count (loge scale) and baseline weight (loge scale) as fixed effects.
- Visit (Day 3, Day 5, Day 10, Day 29, Day 57 and Day 85) and injection site (upper arm, abdomen and thigh) will be fitted as categorical fixed effects variables.
- Treatment-by-visit and baseline blood eosinophil count-by-visit interaction effects will be included in the model as fixed effects.
- Each test treatment (liquid formulation from the autoinjector or safety syringe) will be compared to the reference (reconstituted lyophilised powder from the vial) at each visit.
- The MIXED procedure in SAS will be used with the following options:-

#### **Blood Eosinophil Analyses**

- The Kenward and Roger method (DDFM = KR) for approximating the denominator degrees of freedom to correct for bias in the estimated variance-covariance matrix.
- REPEATED statement with TYPE=UN to specify an unstructured covariance structure for the R matrix.
- The OBSMARGIN option on the LSMEANS statement in order to compute the adjusted geometric means with weights proportional to the input data set.

## **Model Checking & Diagnostics**

- The normality assumption will be examined by obtaining box plots and normal probability plots
  of the studentized marginal residuals at each visit.
- If the model fails to converge, alternative correlation structures will be considered.

#### **Model Results Presentation**

For each visit (Day 3, Day 5, Day 10, Day 29, Day 57 and Day 85):-

- Summary statistics for the ratio to baseline blood eosinophil count.
- Model adjusted geometric mean ratio to baseline blood eosinophils for each treatment group and standard error (log<sub>e</sub> scale).
- Point estimates and associated two-sided 95% confidence intervals for the ratio of each of the
  test treatments to the reference treatment (obtained by back-transforming estimates and 95%
  Cls for the treatment differences from the repeated measures statistical model on the loge
  scale).

## 10.2. User/Device Errors

Summaries of the user/device errors will be based on the "All Treated" population.

Any user/device errors reported on the 'Injection Assessment' page in the eCRF will be summarised and listed by test treatment. Details of the data displays to be presented are given in Appendix 10: List of Data Displays.

## 11. REFERENCES

GlaxoSmithKline Document Number 2016N275057\_02 Study ID 204958. Clinical Protocol for Study 204958: An open label, randomised, three arm, single dose, multicentre, parallel group study in healthy subjects to compare the pharmacokinetics of subcutaneous mepolizumab when delivered as a liquid drug product in a safety syringe or an auto injector with a reconstituted lyophilised drug product from a vial. Report Date 17-NOV-2016.

# 12. APPENDICES

| Section | Appendix |
|---|---|
| RAP Section 5 | : General Considerations for Data Analyses & Data Handling Conventions |
| Section 12.1 | Appendix 1: Time & Events |
| Section 12.2 | Appendix 2: Treatment States and Phases |
| Section 12.3 | Appendix 3: Data Display Standards & Handling Conventions |
| | Study Treatment & Injection Site Descriptors |
| | Baseline Definition & Derivations |
| | Reporting Process & Standards |
| Section 12.4 | Appendix 4: Derived and Transformed Data |
| | General |
| | Study Population |
| | Pharmacokinetics |
| | Safety |
| | Blood Eosinophils |
| Section 12.5 | Appendix 5: Premature Withdrawals & Handling of Missing Data |
| Section 12.6 | Appendix 6: Values of Potential Clinical Importance |
| Section 12.7 | Appendix 7: Multicenter Studies |
| Section 12.8 | Appendix 8: Examination of Covariates, Subgroups & Other Strata |
| Other RAP App | pendices |
| Section 12.9 | Appendix 9: Abbreviations & Trade Marks |
| Section 12.10 | Appendix 10: List of Data Displays |
| Section 12.11 | Appendix 11: Example Mock Shells for Data Displays |

# 12.1. Appendix 1: Time & Events

## 12.1.1. Protocol Defined Time & Events

| | | Trea | tment | Period | 1 [Day | <b>s</b> ] | | | | | | | | | | | | | Notes: |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Procedure | Screening<br>(up to 30<br>days prior<br>to Day 1) | Day -1 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 15 | 22 | 29 | 43 | 57 | 85<br>(FUP/EW) | |
| Informed consent | X | | | | | | | | | | | | | | | | | | |
| Inclusion and exclusion criteria | Х | Х | | | | | | | | | | | | | | | | | |
| Demography | Х | | | | | | | | | | | | | | | | | | |
| Full physical exam including height <sup>1</sup> and weight <sup>2</sup> | Х | X | | | | | | | | | | | | | | | | Х | <sup>1</sup> Height only at<br>screening<br><sup>2</sup> Weight collected only<br>at day -1 |
| Medical history (includes substance usage) Including Cardiovascular medical history/risk factors | х | | | | | | | | | | | | | | | | | | |
| Alcohol test | Х | Х | | | | | | | | | | | | | | | | | Alcohol measured in<br>Serum |
| Drug Screen | Х | Х | | | | | | | | | | | | | | | | | Serum or Urine drug screen |
| Urine Cotinine test | Х | Х | | | | | | | | | | | | | | | | | Tobacco |

| | | Treat | ment | Period ' | 1 [Days] | | | | | | | | | | | | | | Notes: |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Procedure | Screening<br>(up to 30<br>days prior<br>to Day 1) | Day -1 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 15 | 22 | 29 | 43 | 57 | 85<br>(FUP/EW) | |
| Past and current medical conditions | Х | | | | | | | | | | | | | | | | | | |
| Pregnancy test | Х | Х | | | | | | | | | | | | | Х | | | Х | All pregnancy tests will be performed in urine. |
| Laboratory<br>assessments<br>including<br>haematology,<br>chemistry and<br>urinalysis | х | Х | | | | | Х | | | | | | | | | | | Х | Includes Liver chemistry |
| HIV, Hep B and<br>Hep C screen | х | | | | | | | | | | | | | | | | | | If test otherwise<br>performed within 3<br>months prior to first<br>dose of study<br>treatment, testing at<br>screening is not<br>required |
| Immunogenicity | Х | | <b>X</b> <sup>3</sup> | | | | | | | | | | | | Х | Х | | Х | <sup>3</sup> Day 1 Predose.<br>Including binding and<br>neutralising antibody |
| 12-lead ECG | Х | | Χ | | | | | | | | | | | | | | | Х | Day 1 – Predose |
| Vital signs | Х | Х | X <sup>4</sup> | Х | Х | Х | Х | Х | Х | | | | | | | Χ | | Х | <sup>4</sup> Day 1 – Predose |

| | | Treat | ment | Period | 1 [Days] | ] | | | | | | | | | | | | | Notes: |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Procedure | Screening<br>(up to 30<br>days prior<br>to Day 1) | Day -1 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 15 | 22 | 29 | 43 | 57 | 85<br>(FUP/EW) | |
| Parasite screening | <b>X</b> 5 | | | | | | | | | | | | | | | | | | <sup>5</sup> Only required in high risk countries or for subjects who have visited high risk countries in the past six months. Sites should use local laboratories |
| Randomisation | | | Χ | | | | | | | | | | | | | | | | |
| Study Treatment | | | х | | | | | | | | | | | | | | | | Complete either the autoinjector or the safety syringe functionality assessment when applicable |
| AE review | | Х | <b>←</b> = | ===== | ===== | ===== | :===== | ===== | ===== | ==== | === | ==== | ==== | ==== | ===== | :==== | :===: | | Including local<br>injection site reactions<br>and systemic<br>reactions<br>Collected from day -1<br>to Day 85 |
| SAE review | Х | х | ←======> | | | | | | Including local injection site reactions and systemic reactions Collected from screening to Day 85 | | | | | | | | | | |
| Concomitant medication review | Х | Χ | <b>←=</b> : | ===== | ===== | | ===== | ===== | ===== | ==== | | ==== | | ==== | | | | <del>-</del> | Collected from screening to Day 85 |

| | Screening<br>(up to 30<br>days prior<br>to Day 1) | Treatment Period 1 [Days] | | | | | | | | | | | | | | Notes: | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Procedure | | Day -1 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 15 | 22 | 29 | 43 | 57 | 85<br>(FUP/EW) | |
| Blood Samples for PK | | | X6 | Х | Х | Х | Х | X | Х | Х | Х | Х | Х | Х | X | Х | Х | Х | <sup>6</sup> Day 1 – Predose, 2h<br>& 8h Postdose |
| Blood samples for PD (blood eosinophils) | | | X <sup>7</sup> | | Х | | Х | | | | | Х | | | Х | | Х | Х | <sup>7</sup> Day 1 – Predose |
| Autoinjector and safety syringe user/device error assessment- | | | Х | | | | | | | | | | | | | | | | HCP reported. |
| Follow up (FUP) | | | | | | | | | | | | | | | | | | Χ | |

# 12.2. Appendix 2: Treatment States and Phases

## 12.2.1. Treatment Phases

Assessments and events will be classified according to the time of occurrence relative to the dose of study treatment.

## 12.2.1.1. Treatment Phases for Adverse Events

| Treatment State | Definition |
|---|---|
| Pre-Treatment | AE start date < Mepolizumab dosing date |
| On-Treatment | <ul> <li>Mepolizumab dosing date ≤ AE start date ≤ Mepolizumab dosing date + 28 days</li> <li>Any adverse event with missing start date will be assumed to be "On-Treatment".</li> </ul> |
| | <ul> <li>Any adverse event with partial start date will be assumed to be "On-Treatment"<br/>unless there is evidence to the contrary (e.g. month/year of onset is present<br/>and is earlier than the month/year of the dose of study treatment).</li> </ul> |
| Post-Treatment | AE start date > Mepolizumab dosing date + 28 days |

# 12.3. Appendix 3: Data Display Standards & Handling Conventions

## 12.3.1. Study Treatment & Injection Site Descriptors

Separate descriptors for treatment group and injection site will be assigned as follows:-

| | Treatment Group Descriptions <sup>[1]</sup> | | |
|---|---|---|---|
| | RandAll NG | Data Displays for Reporting | |
| Code | Description | Treatment Group Description | Order [2] |
| A1 | Liquid auto injector - abdomen | Liquid Autoinjector | 2 |
| A2 | Liquid auto injector – arm | Liquid Autoinjector | 2 |
| A3 | Liquid auto injector – thigh | Liquid Autoinjector | 2 |
| S1 | Liquid safety syringe - abdomen | Liquid Safety Syringe | 3 |
| S2 | Liquid safety syringe – arm | Liquid Safety Syringe | 3 |
| S3 | Liquid safety syringe – thigh | Liquid Safety Syringe | 3 |
| R1 | Reconstituted lyophilised – abdomen | Lyophilised Vial | 1 |
| R2 | Reconstituted lyophilised – arm | Lyophilised Vial | 1 |
| R3 | Reconstituted lyophilised – thigh | Lyophilised Vial | 1 |

#### NOTES:

- 1. For summaries of safety data, a "Total Liquid" column will present the combined results from the liquid autoinjector and liquid safety syringe, and a "Total" column will present the combined results across all 3 randomised treatment groups.
- 2. Order represents treatments being presented in TFL, as appropriate.

| | Injection Site Descriptions | | |
|---|---|---|---|
| | RandAll NG | Data Displays for Reporti | ng |
| Code | Description | Injection Site Description | Order [1] |
| A1 | Liquid auto injector - abdomen | Abdomen | 1 |
| A2 | Liquid auto injector – arm | Arm | 2 |
| A3 | Liquid auto injector – thigh | Thigh | 3 |
| S1 | Liquid safety syringe - abdomen | Abdomen | 1 |
| S2 | Liquid safety syringe – arm | Arm | 2 |
| S3 | Liquid safety syringe – thigh | Thigh | 3 |
| R1 | Reconstituted lyophilised – abdomen | Abdomen | 1 |
| R2 | Reconstituted lyophilised – arm | Arm | 2 |
| R3 | Reconstituted lyophilised – thigh | Thigh | 3 |

#### NOTES:

1. Order represents treatments being presented in TFL, as appropriate.

#### 12.3.2. Baseline Definition & Derivations

#### 12.3.2.1. Baseline Definitions

- Baseline will be defined for all subjects in the 'All Treated Subjects" population.
- The baseline values for each assessment will be the latest available assessment prior to receiving the single dose of mepolizumab.

## 12.3.2.2. Derivations and Handling of Missing Baseline Data

| Definition | Reporting Details |
|---|---|
| Change from Baseline | = Post-Dose Visit Value – Baseline |
| % Change from Baseline | = 100 x [(Post-Dose Visit Value – Baseline) / Baseline] |
| Ratio to Baseline | = Visit Value / Baseline |

#### NOTES:

- Unless otherwise specified, the baseline definitions specified in Section 12.3.2.1 will be used for derivations for endpoints / parameters and indicated on summaries and listings.
- Unless otherwise stated, if baseline data is missing no derivation will be performed and will be set to missing.

## 12.3.3. Reporting Process & Standards

| Reporting Process | Reporting Process |
|---|---|
| Software | Software |
| The currently supported versions of SAS software will be used. | |
| Reporting Area | |
| HARP Server | : uk1salx00175 |
| HARP Area | : sb240563/mid204958 |
| <b>Analysis Datasets</b> | |
| <ul> <li>Analysis datasets</li> </ul> | Analysis datasets will be created according to CDISC standards. |
| <ul> <li>For creation of ADaM datasets (ADCM/ADAE), the same version of dictionary datasets will be<br/>implemented for conversion from SI to SDTM.</li> </ul> | |
| Generation of RTF F | Files |

## **Reporting Standards**

#### General

- The current GSK Integrated Data Standards Library (IDSL) will be applied for reporting, unless otherwise stated:
  - 4.03 to 4.23: General Principles
  - 5.01 to 5.08: Principles Related to Data Listings

RTF files will be generated for final reporting effort.

- o 6.01 to 6.11: Principles Related to Summary Tables
- 7.01 to 7.13: Principles Related to Graphics
- Listings will include treatment and injection site (see Section 12.3.1).

#### **Reporting Standards**

#### **Formats**

 The reported precision (decimal places) will follow the IDSL statistical principles but may be adjusted to a clinically interpretable number of DPs.

#### **Planned and Actual Time**

- Reporting for tables, figures and formal statistical analyses :
  - Actual time relative to dosing will be used for individual subject plasma concentration-time figures and for derivation of PK parameters.
  - Planned time relative to dosing will be used in all other figures, summaries, statistical analyses and calculation of any derived parameters.
  - The impact of any major deviation from the planned assessment times and/or scheduled visit days on the analyses and interpretation of the results will be assessed as appropriate.
- Reporting for Data Listings:
  - Planned and actual time relative to study drug dosing will be shown in listings (Refer to IDSL Statistical Principle 5.05.1).
  - Unscheduled or unplanned readings will be presented within the subject's listings.
- Visits outside the protocol defined time-windows (i.e. recorded as protocol deviations) will be included in listings, summaries and statistical analyses.

#### **Unscheduled Visits**

- Data recorded at an unscheduled visit will be re-assigned to the closest nominal visit at which
  collection of data was scheduled, unless information already exists at that visit. Unscheduled
  data re-assigned to a scheduled visit will be reported in summary tables and figures.
  Unscheduled data that is not re-assigned to a scheduled visit will not be included in summary
  tables or figures.
- All unscheduled visits will be included in listings and individual subject figures.

| Descriptive Summary Statistics | |
|---|---|
| Continuous Data | Refer to IDSL Statistical Principle 6.06.1 |
| Categorical Data | N, n, frequency, % |
| Reporting of Pharm | Reporting of Pharmacokinetic Concentration Data |
| Descriptive<br>Summary Statistics<br>(All Parameters) | N, n, no. imputed, mean, 95% CI for mean, standard deviation, minimum, median and maximum will be reported. Assign zero to NQ values (Refer to GUI_51487 for further details) |

| Reporting Standard | Reporting Standards |
|---|---|
| Reporting of Pharm | acokinetic Parameters |
| Descriptive Summary Statistics (All parameters) | N, n, mean, 95% CI for mean, standard deviation, minimum, median and maximum will be reported. |
| Log-Normal<br>Parameters | Cmax, AUC(0-∞), AUC(0-t), AUC(0-week4), CL/F, Vd/F, λz, t½, %AUCextrapolated |
| Additional Descriptive Summary Statistics (Log-Normal parameters) | N, n, geometric mean, 95% CI of geometric mean, standard deviation (SD) of logged data and coefficient of variation (CVb (%)) will be reported. $ \text{CV}_b \text{ (\%)} = \sqrt{(\text{exp}(\text{SD}^2) - 1) * 100} $ (SD = SD of log transformed data) |
| Parameters to be listed only | Number of points used to determine $\lambda z$ |
| Graphical Displays | |
| Refer to IDSL Statistical Principals 7.01 to 7.13. | |

## 12.4. Appendix 4: Derived and Transformed Data

#### 12.4.1. **General**

#### Multiple Measurements at One Time Point

- May arise when unscheduled visits are re-assigned to a nominal visit (see Section 12.3.3). If
  there is data at the nominal visit, the nominal visit data will be used in the summary tables and
  figures. All assessments will be listed.
- Subjects having both High and Low values for Normal Ranges at any post-baseline visits for safety parameters will be counted in both the High and Low categories of "Any visit postbaseline" row of related summary tables. This will also be applicable to relevant Potential Clinical Importance summary tables.

#### **Study Day**

Calculated as the number of days from dosing date for mepolizumab:

Ref Date = Missing  $\rightarrow$  Study Day = Missing

Ref Date < Mepolizumab dosing date → Study Day = Ref Date – Mepolizumab dosing date

Ref Data ≥ Mepolizumab dosing date → Study Day = Ref Date – Mepolizumab dosing date + 1

#### 12.4.2. Study Population

## **Demographics**

#### Age

- GSK standard IDSL algorithms will be used for calculating age where birth day and month will be imputed '30th June'.
- Birth date will be presented in listings as 'YYYY'.
- Age will be calculated relative to the date of the screening visit (Visit 1).

#### **Body Mass Index (BMI)**

• Calculated as Weight (kg) / [Height (m)<sup>2</sup>]

#### **Extent of Exposure**

As this is a single dose study, exposure data will be listed only.

#### 12.4.3. Pharmacokinetics

Derivation of pharmacokinetic parameters is detailed in Section 7.3.

## 12.4.4. Safety

#### **Adverse Events**

## **Drug Related AEs**

AEs with relationship marked 'YES' or relationship missing.

#### AE Time Since First Dose (Days)

• If AE start date < Mepolizumab dosing date then

Time since first dose = Mepolizumab dosing date - AE start date

If AE start date ≥ Mepolizumab dosing date then

Time since first dose = AE start date – Mepolizumab dosing date +1

Missing if AE start date or mepolizumab dosing date is missing.

## AE Duration (Days)

- AE end date AE start date + 1
- Missing if AE start date or end date is missing.

#### AEs of Special Interest

See Section 8.1.1

## 12.4.5. Blood Eosinophils

See Section 10.1.1 for handling of non-detectable blood eosinophil values of 0 GI/L.

# 12.5. Appendix 5: Premature Withdrawals & Handling of Missing Data

## 12.5.1. Premature Withdrawals

| Element | Reporting Detail |
|---|---|
| General | <ul> <li>Subject study completion is defined as completion of assessments on Day 85.</li> <li>Withdrawn subjects will not be replaced in the study.</li> <li>All available data from subjects who were withdrawn from the study will be listed</li> </ul> |
| | and all available planned data will be included in summary tables and figures, unless otherwise specified. |
| Screen<br>Failures | <ul> <li>A subject will be assigned a subject number at the time when the informed<br/>consent form (ICF) is signed.</li> </ul> |
| | <ul> <li>A subject who is assigned a subject number, but is never subsequently<br/>randomised will be considered a screen failure.</li> </ul> |

# 12.5.2. Handling of Missing Data

| Element | Reporting Detail |
|---|---|
| General | <ul> <li>Analysis will be performed on all available data and no imputation will be performed for missing data</li> <li>Missing data occurs when any requested data is not provided, leading to blank fields on the collection instrument. These data will be indicated by the use of a "blank" in subject listing displays, unless all data for a specific visit are missing in which case the data is excluded from the listing.</li> <li>Data below the limit of quantification (BLQ) is not missing data and must be displayed as such and included in all listings and summaries.</li> </ul> |
| Outliers | Any subjects excluded from the summaries and/or statistical analyses because their values are considered outliers will be documented along with the reason for exclusion in the clinical study report. |

# 12.5.2.1. Handling of Missing and Partial Dates

| Element | Reporting Detail |
|---|---|
| General | Partial dates will be displayed as captured in subject listing displays. |
| Adverse<br>Events | <ul> <li>Any partial dates for adverse events will be raised to data management. If the full date cannot be ascertained, the following assumptions will be made: <ul> <li>If the partial date is a start date, a '01' will be used for the day and 'Jan' will be used for the month.</li> </ul> </li> </ul> |
| | <ul> <li>However, if this imputation results in a date prior to the first dose of<br/>mepolizumab and the event could possibly have occurred during treatment<br/>from the partial information, then the date of the first dose of mepolizumab<br/>will be assumed to be the start date.</li> </ul> |
| | <ul> <li>The event will then be considered to start on-treatment (worst case).</li> <li>If the partial date is a stop date, a '28/29/30/31' will be used for the day (dependent on the month and year) and 'Dec' will be used for the month.</li> </ul> |
| | Completely missing start or end dates will remain missing, with no imputation applied. Consequently, time to onset and duration of such events will be missing. Adverse events with completely missing start dates will be considered to start on-treatment (worst case). |
| | The recorded partial date will be displayed in listings. |
# 12.6. Appendix 6: Values of Potential Clinical Importance

### 12.6.1. Laboratory Values of Potential Clinical Concern

| Haematology | | | | |
|---|---|---|---|---|
| Laboratory Parameter Units Age Clinical Concern Range | | | | |
| | | Category | Low Flag (< x) | High Flag (>x) |
| Hematocrit | Ratio of 1 | 12+ | 0.201 | 0.599 |
| Hemoglobin | G/L | 12+ | 71 | 199 |
| Platelet Count | GI/L | 1+ | 31 | 1499 |
| While Blood Cell Count (WBC) | GI/L | 12+ | 1.1 | |

| Clinical Chemistry | | | | |
|---|---|---|---|---|
| Laboratory Parameter | Units | Age | Clinical Concern Range | |
| | | Category | Low Flag (< x) | High Flag (>x) |
| ALT | U/L | 3-12 | | >143 (and Total<br>Bilirubin >43) |
| | U/L | 13+ | | >239 (and Total<br>Bilirubin >43) |
| Calcium | mmol/L | 3+ | 1.50 | 3.24 |
| Glucose | mmol/L | 1+ | 2.2 | 27.8 |
| Phosphorus, Inorg | mmol/L | 3+ | 0.32 | |
| Potassium | mmol/L | 3+ | 2.8 | 6.5 |
| Sodium | mmol/L | 0+ | 120 | 160 |

| Possible Hy's Law Cases | | | |
|---|---|---|---|
| Laboratory Parameter | Units | Category | Clinical Concern Range |
| ALT, Bilirubin | | | ALT ≥ 3xULN and Bilirubin ≥ 2xULN (>35% direct) |
| ALT, INR | | | ALT ≥ 3xULN and INR > 1.5 |

### 12.7. Appendix 7: Multicenter Studies

- This study will be conducted in 3 centres attributed to a single contract research organisation (CRO).
- The randomisation for this study is allocated centrally.
- Centre will not be included as a covariate in the statistical analyses for this study.

# 12.8. Appendix 8: Examination of Covariates, Subgroups & Other Strata

### 12.8.1. Handling of Covariates

• Baseline body weight, on log<sub>e</sub> scale will be included as a covariate in all statistical analyses. For analyses where a baseline value (of the analysis variable) is available this will also be included in the statistical analysis. These covariates will be included as fixed effects in the statistical model.

### 12.8.2. Handling of Subgroups

- Pharmacokinetic concentrations and parameters will be summarised by baseline weight category (<70 kg, 70-<80 kg and ≥80 kg) and injection site see Section 7.2 and Section 7.3. No formal statistical analysis of these subgroups is planned.
- No subgroup analyses are planned for any other study endpoints.

# 12.9. Appendix 9: Abbreviations & Trade Marks

### 12.9.1. Abbreviations

| Abbreviation | Description |
|--------------|--------------------------------------------------|
| ADA | Anti-Drug Antibody |
| ADaM | Analysis Data Model |
| AE | Adverse Event |
| A&R | Analysis and Reporting |
| BLQ | Below the Limit of Quantification |
| CDISC | Clinical Data Interchange Standards Consortium |
| CI | Confidence Interval |
| CPMS | Clinical Pharmacology Modelling & Simulation |
| CS | Clinical Statistics |
| CSR | Clinical Study Report |
| CTR | Clinical Trial Register |
| $CV_b$ | Coefficient of Variation (Between) |
| DOB | Date of Birth |
| DP | Decimal Places |
| eCRF | Electronic Case Record Form |
| GUI | Guidance |
| ICH | International Conference on Harmonisation |
| IDSL | Integrated Data Standards Library |
| IMMS | International Modules Management System |
| IP | Investigational Product |
| PCI | Potential Clinical Importance |
| PD | Pharmacodynamic |
| PDMP | Protocol Deviation Management Plan |
| PK | Pharmacokinetic |
| QC | Quality Control |
| QTcF | Frederica's QT Interval Corrected for Heart Rate |
| QTcB | Bazett's QT Interval Corrected for Heart Rate |
| RAP | Reporting & Analysis Plan |
| SAC | Statistical Analysis Complete |
| SDL | Source Data Lock |
| SDTM | Study Data Tabulation Model |
| SOP | Standard Operation Procedure |
| TA | Therapeutic Area |
| TFL | Tables, Figures & Listings |
| GSK | GlaxoSmithKline |

### 12.9.2. Trademarks

| Trademarks of the GlaxoSmithKline |
|-----------------------------------|
| Group of Companies |

NONE

# Trademarks not owned by the GlaxoSmithKline Group of Companies

Phoenix

SAS

# 12.10. Appendix 10: List of Data Displays

# 12.10.1. Study Population Tables

| Study F | Study Population Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 6.1 | ASE | TAB_POP1 | Summary of Study Populations by Treatment | | SAC |
| 6.2 | Randomised | TAB_POP2 | Summary of Study Populations By Treatment and Injection Site | | SAC |
| 6.3 | ASE | ES6 | Summary of Screen Failures | | SAC |
| 6.4 | ASE | NS1 | Summary of Number of Subjects by Country and Site, by Treatment | "Not Treated" column should be added to include subjects who were not randomised, or randomised subjects who did not receive treatment. | SAC |
| 6.5 | ASE | NS1 | Summary of Number of Subjects by Country and Site, by Treatment and Injection Site | "Not Treated" column should be added to include subjects who were not randomised, or randomised subjects who did not receive treatment. | SAC |
| 6.6 | All Treated | ES1 | Summary of Subject Disposition by Treatment | | SAC |
| 6.7 | All Treated | DV1 | Summary of Important Protocol Deviations by Treatment | | SAC |
| 6.8 | All Treated | DM1 | Summary of Demographic Characteristics by Treatment | | SAC |
| 6.9 | All Treated | DM5 | Summary of Race and Racial Combinations by Treatment | | SAC |
| 6.10 | ASE | DM11 | Summary of Age Ranges by Treatment | "Not Treated" column should be added to include subjects who were not randomised, or randomised subjects who did not receive treatment. | SAC |
| 6.11 | All Treated | MH1 | Summary of Past Medical Conditions by Treatment | | SAC |
| 6.12 | All Treated | MH1 | Summary of Current Medical Conditions by Treatment | | SAC |

| Study F | Study Population Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 6.13 | All Treated | FH1 | Summary of Family History of Cardiovascular Risk Factors by Treatment | | SAC |
| 6.14 | All Treated | SU1 | Summary of Smoking History by Treatment | Smoking status (current/former/never) only | SAC |

# 12.10.2. Pharmacokinetic Figures

| Pharma | Pharmacokinetic : Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| PK Con | centration | | | | |
| 7.1 | PK | PK16a | Individual Plasma Mepolizumab Concentration-Time Plots (Linear and Semi-Log) by Subject | Actual body weight category, treatment, injection site and subject number as byline. | SAC |
| 7.2 | PK | PK26 | Individual Plasma Mepolizumab Concentration-Time Plots (Linear and Semi-Log) by Treatment | Treatment as by-line. All subjects receiving the treatment on the same graph ("spaghetti" plot). | SAC |
| 7.3 | PK | PK17 | Mean Plasma Mepolizumab Concentration-Time Plots by<br>Treatment (Linear and Semi-Log) | | SAC |
| 7.4 | PK | PK18 | Median Plasma Mepolizumab Concentration-Time Plots by Treatment (Linear and Semi-Log) | | SAC |
| 7.5 | PK | PK17 | Mean Plasma Mepolizumab Concentration-Time Plots by<br>Treatment and Injection Site (Linear and Semi-Log) | | SAC |

| Pharma | acokinetic : Fig | ures | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 7.6 | PK | PK18 | Median Plasma Mepolizumab Concentration-Time Plots by<br>Treatment and Injection Site (Linear and Semi-Log) | | SAC |
| 7.7 | PK | PK17 | Mean Plasma Mepolizumab Concentration-Time Plots by Baseline Body Weight Category and Treatment (Linear and Semi-Log) | Use actual body weight category | SAC |
| 7.8 | PK | PK18 | Median Plasma Mepolizumab Concentration-Time Plots by Baseline Body Weight Category and Treatment (Linear and Semi-Log) | Use actual body weight category | SAC |
| 7.9 | PK | PK17 | Mean Plasma Mepolizumab Concentration-Time Plots by Baseline Body Weight Category, Treatment and Injection Site (Linear and Semi-Log) | Actual body weight category as by-line. | SAC |
| 7.10 | PK | PK18 | Median Plasma Mepolizumab Concentration-Time Plots by Baseline Body Weight Category, Treatment and Injection Site (Linear and Semi-Log) | Actual body weight category as by-line. | SAC |
| PK Para | ameter | | | | |
| 7.11 | PK | FIG_PK1 | Individual Subject (+Geometric Mean and 95% CI) Derived Plasma Mepolizumab PK Parameters by Treatment | AUC(0-inf), AUC(0-t) and Cmax only | SAC |
| 7.12 | PK | FIG_PK2 | Individual Subject (+Geometric Mean and 95% CI) Derived Plasma Mepolizumab PK Parameters by Treatment and Injection Site | AUC(0-inf), AUC(0-t) and Cmax only | SAC |
| 7.13 | PK | FIG_PK3 | Individual Subject (+Geometric Mean and 95% CI) Derived Plasma Mepolizumab PK Parameters by Baseline Body Weight Category and Treatment | AUC(0-inf), AUC(0-t) and Cmax only Use actual body weight category. | SAC |

| Pharma | Pharmacokinetic : Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 7.14 | PK | FIG_PK4 | Individual Subject (+Geometric Mean and 95% CI) Derived Plasma Mepolizumab PK Parameters by Baseline Body Weight Category, Treatment and Injection Site | AUC(0-inf), AUC(0-t) and Cmax only. Use actual body weight category. | SAC |
| 7.15 | PK | FIG_PK5 | Adjusted Geometric Means and Treatment Ratios (90% CI) for Primary Analysis of Derived Plasma Mepolizumab PK Parameters | AUC(0-inf), AUC(0-t) and Cmax only | SAC |

### 12.10.3. Pharmacokinetic Tables

| Pharma | Pharmacokinetic : Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| PK Con | PK Concentration | | | | |
| 7.1 | PK | PK01 | Summary of Plasma Mepolizumab Concentration-Time Data by Treatment | Treatment as by-line. | SAC |
| 7.2 | PK | PK01 | Summary of Plasma Mepolizumab Concentration-Time Data by Treatment and Injection Site | Treatment and injection site as by-line. | SAC |
| 7.3 | PK | PK01 | Summary of Plasma Mepolizumab Concentration-Time Data by Baseline Body Weight Category and Treatment | Use actual body weight category. | SAC |
| 7.4 | PK | PK01 | Summary of Plasma Mepolizumab Concentration-Time Data by Baseline Body Weight Category, Treatment and Injection Site | Use actual body weight category. Body weight category, treatment and injection site as by-line. | SAC |

| Pharma | Pharmacokinetic : Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| PK Par | ameter | | | | |
| 7.5 | PK | PK03 | Summary of Untransformed Derived Plasma Mepolizumab Pharmacokinetic Parameters by Treatment | Cmax, AUC(0-∞), AUC(0-t), AUC(0-week4), CL/F, Vd/F, λz, t½, %AUCextrapolated, tmax, tlast | SAC |
| 7.6 | PK | PK05 | Summary of Log-transformed Derived Plasma Mepolizumab Pharmacokinetic Parameters by Treatment | Cmax, AUC(0-∞), AUC(0-t), AUC(0-week4), CL/F, Vd/F, λz, t½, %AUCextrapolated | SAC |
| 7.7 | PK | PK03 | Summary of Untransformed Derived Plasma Mepolizumab Pharmacokinetic Parameters by Treatment and Injection Site | Parameter as by-line. See Table 7.5 for list of parameters. | SAC |
| 7.8 | PK | PK05 | Summary of Log-transformed Derived Plasma Mepolizumab Pharmacokinetic Parameters by Treatment and Injection Site | Parameter as by-line. See Table 7.6 for list of parameters. | SAC |
| 7.9 | PK | PK03 | Summary of Untransformed Derived Plasma Mepolizumab Pharmacokinetic Parameters by Baseline Body Weight Category and Treatment | Use actual body weight category. Parameter as by-line. See Table 7.5 for list of parameters. | SAC |
| 7.10 | PK | PK05 | Summary of Log-transformed Derived Plasma Mepolizumab Pharmacokinetic Parameters by Baseline Body Weight Category and Treatment | Use actual body weight category. Parameter as by-line. See Table 7.6 for list of parameters. | SAC |
| 7.11 | PK | PK03 | Summary of Untransformed Derived Plasma Mepolizumab Pharmacokinetic Parameters by Baseline Body Weight Category, Treatment and Injection Site | Use actual body weight category. Parameter and body weight category as by-line. See Table 7.5 for list of parameters. | SAC |

| Pharmacokinetic : Tables | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 7.12 | PK | PK05 | Summary of Log-transformed Derived Plasma Mepolizumab Pharmacokinetic Parameters by Baseline Body Weight Category, Treatment and Injection Site | Use actual body weight category. Parameter and body weight category as by-line. See Table 7.6 for list of parameters. | SAC |
| 7.13 | PK | TAB_PK1 | Summary of Statistical Analysis of Derived Plasma Mepolizumab AUC(0-inf), AUC(0-t) and Cmax | | SAC |

### 12.10.4. Safety Tables

### Programming Note:

For all safety tables, five treatment groups should appear as follows: Lyophilised Vial, Liquid Autoinjector, Liquid Safety Syringe, Total Liquid and Total.

| Safety : | Safety : Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Advers | e Events | | | | |
| 8.1 | All Treated | AE1 | Summary of All On-Treatment Adverse Events by System Organ Class and Preferred Term | | SAC |
| 8.2 | All Treated | AE1 | Summary of All Post-Treatment Adverse Events by System<br>Organ Class and Preferred Term | | SAC |
| 8.3 | All Treated | AE3 | Summary of Common (>=3% Incidence [1]) On-Treatment Adverse Events by Overall Frequency | Add footnote as follows:- [1] AEs with >=3% Incidence in either the Total Liquid or Lyophilised Vial treatment groups are presented. | SAC |
| 8.4 | All Treated | AE15 | Summary of Common (>=3% Incidence[1]) On-Treatment Adverse Events by Preferred Term (Number of Subjects and Occurrences) | Add footnote as follows:- [1] AEs with >=3% Incidence in either the Total Liquid or Lyophilised Vial treatment groups are presented. | SAC |
| 8.5 | All Treated | AE5A | Summary of All On-Treatment Adverse Events by Maximum Intensity by System Organ Class and Preferred Term | | SAC |
| 8.6 | All Treated | AE1 | Summary of All Drug-Related Adverse Events by System Organ Class and Preferred Term | | SAC |

| Safety | Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 8.7 | All Treated | AE5A | Summary of All Drug-Related Adverse Events by Maximum Intensity by System Organ Class and Preferred Term | | SAC |
| 8.8 | All Treated | AE1 | Summary of On-Treatment Adverse Events by Highest Post-<br>Baseline Binding Antibody Result | Add in row with n in each binding antibody result category (negative, Transient positive, Persistent positive). See Section 9 for derivation of highest post-baseline binding antibody result. | SAC |
| 8.9 | All Treated | AE3 | Summary of All Adverse Events Leading to Withdrawal from the Study by Overall Frequency | | SAC |
| 8.10 | All Treated | AE1 | Summary of Adverse Events Reported on the Day of Dosing by System Organ Class and Preferred Term | | SAC |
| 8.11 | All Treated | AE7 | Listing of Subject Numbers for Individual On-Treatment Adverse Events | | SAC |
| 8.12 | All Treated | AE2 | Listing of Relationship of Adverse Event, System Organ Classes, Preferred Terms and Verbatim Text | | SAC |
| Serious | Adverse Ever | nts | | , | |
| 8.13 | All Treated | AE3 | Summary of Fatal Serious Adverse Events by Overall Frequency | | SAC |
| 8.14 | All Treated | AE3 | Summary of Drug-Related Fatal Serious Adverse Events by Overall Frequency | | SAC |
| 8.15 | All Treated | AE1 | Summary of All On-Treatment Serious Adverse Events by<br>System Organ Class and Preferred Term | | SAC |

| Safety : | Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 8.16 | All Treated | AE16 | Summary of All On-Treatment Serious Adverse Events by<br>System Organ Class and Preferred Term (Number of Subjects<br>and Occurrences) | | SAC |
| 8.17 | All Treated | AE1 | Summary of All Post-Treatment Serious Adverse Events by System Organ Class and Preferred Term | | SAC |
| 8.18 | All Treated | AE1 | Summary of All Pre-Treatment Serious Adverse Events by<br>System Organ Class and Preferred Term | | SAC |
| 8.19 | All Treated | AE1 | Summary of All Drug-Related Serious Adverse Events by System Organ Class and Preferred Term | | SAC |
| Advers | e Events of Sp | ecial Interest | | • | |
| 8.20 | All Treated | AE1 | Summary of On-Treatment Adverse Events Reported by the Investigator as Meeting the Criteria for Anaphylaxis | | SAC |
| 8.21 | All Treated | TAB_S1 | Summary Profile of On-Treatment Adverse Events Reported by the Investigator as Meeting the Criteria for Anaphylaxis | | SAC |
| 8.22 | All Treated | AE1 | Summary of On-Treatment Adverse Events Defined by the Investigator as Systemic Reactions - Allergic (Type I Hypersensitivity) and Other Systemic | | SAC |
| 8.23 | All Treated | TAB_S1 | Summary Profile of On-Treatment Adverse Events Defined by the Investigator as Systemic Reactions - Allergic (Type I Hypersensitivity) and Other Systemic | | SAC |
| 8.24 | All Treated | AE1 | Summary of On-Treatment Adverse Events Defined by the Investigator as Systemic Reactions - Allergic (Type I Hypersensitivity) | | SAC |

| Safety | Safety : Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 8.25 | All Treated | TAB_S1 | Summary Profile of On-Treatment Adverse Events Defined by the Investigator as Systemic Reactions - Allergic (Type I Hypersensitivity) | | SAC |
| 8.26 | All Treated | AE1 | Summary of On-Treatment Adverse Events Defined by the Investigator as Systemic Reactions – Other Systemic | | SAC |
| 8.27 | All Treated | TAB_S1 | Summary Profile of On-Treatment Adverse Events Defined by the Investigator as Systemic Reactions - Other Systemic | | SAC |
| 8.28 | All Treated | AE1 | Summary of On-Treatment Adverse Events Defined by the Investigator as Local Injection Site Reactions | | SAC |
| 8.29 | All Treated | TAB_S1 | Summary Profile of On-Treatment Adverse Events Defined by the Investigator as Local Injection Site Reactions | | SAC |
| 8.30 | All Treated | AE1 | Summary of On-Treatment Adverse Events Categorised as Serious Cardiac, Vascular and Thromboembolic Events | | SAC |
| 8.31 | All Treated | TAB_S1 | Summary Profile of On-Treatment Adverse Events Categorised as Serious Cardiac, Vascular and Thromboembolic Events | | SAC |
| 8.32 | All Treated | AE1 | Summary of On-Treatment Adverse Events Categorised as Serious Ischemic Events | | SAC |
| 8.33 | All Treated | TAB_S1 | Summary Profile of On-Treatment Adverse Events Categorised as Serious Ischemic Events | | SAC |
| 8.34 | All Treated | AE1 | Summary of On-Treatment Adverse Events Categorised as Malignancies | | SAC |

| Safety | : Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 8.35 | All Treated | TAB_S1 | Summary Profile of On-Treatment Adverse Events Categorised as Malignancies | | SAC |
| 8.36 | All Treated | AE1 | Summary of On-Treatment Adverse Events Categorised as Opportunistic Infections | | SAC |
| 8.37 | All Treated | TAB_S1 | Summary Profile of On-Treatment Adverse Events Categorised as Opportunistic Infections | | SAC |
| Labora | tory - Haemato | logy | | | |
| 8.38 | All Treated | LB1 | Summary of Haematology Changes from Baseline by Visit | Include baseline values | SAC |
| 8.39 | All Treated | LB3 | Summary of Haematology Shifts from Baseline Relative to Normal Range by Visit | | SAC |
| 8.40 | All Treated | LB3 | Summary of Haematology Shifts from Baseline Relative to PCI Criteria by Visit | | SAC |
| Labora | tory – Clinical ( | Chemistry | | 1 | - |
| 8.41 | All Treated | LB1 | Summary of Clinical Chemistry Changes from Baseline by Visit | Include baseline values | SAC |
| 8.42 | All Treated | LB3 | Summary of Clinical Chemistry Shifts from Baseline Relative to Normal Range by Visit | | SAC |
| 8.43 | All Treated | LB3 | Summary of Clinical Chemistry Shifts from Baseline Relative to PCI Criteria by Visit | | SAC |

| Safety : | Safety : Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| ECG | | | | | |
| 8.44 | All Treated | EG1 | Summary of ECG Findings by Visit | | SAC |
| 8.45 | All Treated | EG2 | Summary of ECG Values by Visit | | SAC |
| 8.46 | All Treated | EG2 | Summary of Change from Baseline in ECG Values by Visit | Include baseline values | SAC |
| Vital Sig | gns | | | | |
| 8.47 | All Treated | VS1 | Summary of Vital Signs by Visit | | SAC |
| 8.48 | All Treated | VS1 | Summary of Change from Baseline in Vital Signs by Visit | Include baseline values | SAC |

# 12.10.5. Immunogenicity Tables

| Immuno | Immunogenicity : Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 9.1 | All Treated | TAB_S2 | Summary of Binding Antibody by Visit | Include highest post-baseline result. If highest post-baseline result is positive, include summary statistics (minimum, median, maximum) for titre value – see shell. | SAC |
| 9.2 | All Treated | TAB_S2 | Summary of Binding Antibody By Visit – Subjects Without Positive Result Prior to Dosing | Post-Day 1 visits only, plus highest post-baseline result and titre summary | SAC |

| Immund | Immunogenicity : Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 9.3 | All Treated | TAB_S3 | Summary of Neutralising Antibody by Visit | Include highest post-baseline result. If highest post-baseline result is positive, include summary statistics (minimum, median, maximum) for titre value – see shell. | SAC |

# 12.10.6. Exploratory Figures

| Explora | Exploratory : Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Blood E | osinophils | | | | |
| 10.1 | All Treated | FIG_PD1 | Adjusted Geometric Mean (95% CI) Ratio to Baseline Blood Eosinophils by Visit | Adjusted geometric means for each treatment from statistical analysis. | SAC |
| 10.2 | All Treated | FIG_PD2 | Adjusted Treatment Ratios (95% CI) for Ratio to Baseline Blood Eosinophils by Visit | Treatment ratios relative to lyophilised vial formation from statistical analysis. | SAC |

# 12.10.7. Exploratory Tables

| Explora | Exploratory : Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Blood E | osinophils | | | | |
| 10.1 | PD | TAB_PD1 | Summary of Blood Eosinophils (Gl/L) by Visit | | SAC |
| 10.2 | PD | TAB_PD2 | Summary of Ratio to Baseline Blood Eosinophils by Visit | | SAC |
| 10.3 | PD | TAB_PD3 | Summary of Statistical Analysis of Blood Eosinophils Ratio to Baseline | | SAC |
| User/De | User/Device Errors | | | | |
| 10.4 | All Treated | TAB_AI | Summary of Injection Assessment – Liquid Autoinjector | | SAC |
| 10.5 | All Treated | TAB_SS | Summary of Injection Assessment – Liquid Safety Syringe | | SAC |

# 12.10.8. ICH and Other Listings

| ICH an | ICH and Other Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Study | Population | • | | | |
| 1 | ASE | ES7 | Listing of Reasons for Screen Failure | | SAC |
| 2 | Randomised | SP3 | Listing of Subjects Excluded from Any Population | | SAC |
| 3 | All Treated | TA1 | Listing of Randomised and Actual Treatment | | SAC |
| 4 | All Treated | ES2 | Listing of Reasons for Withdrawal | | SAC |
| 5 | All Treated | DV2 | Listing of Important Protocol Deviations | | SAC |
| 6 | All Treated | IE3 | Listing of Subjects with Inclusion/Exclusion Criteria Deviations | | SAC |
| 7 | All Treated | EX3 | Listing of Exposure Data | | SAC |
| 8 | All Treated | DM2 | Listing of Demographic Characteristics | | SAC |
| 9 | All Treated | DM9 | Listing of Race | | SAC |
| 10 | All Treated | MH2 | Listing of Medical Conditions | | SAC |
| 11 | All Treated | FH5 | Listing of Family History | | SAC |
| 12 | All Treated | CM3 | Listing of Concomitant Medications | Include all data collected on the CRF, plus study day for start date | SAC |
| PK Co | ncentration | | | | |
| 13 | PK | PK07 | Listing of Plasma Concentration-Time Data | Actual body weight category, treatment and injection site as by-line. | SAC |
| 14 | PK | PK13 | Listing of Derived Plasma Mepolizumab Phamacokinetic Parameters | Actual body weight category, treatment and injection site as by-line. | SAC |

| ICH and | ICH and Other Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Advers | Adverse Events | | | | |
| 15 | All Treated | AE8 | Listing of All Adverse Events | Add phase: Pre-treatment, on-<br>treatment, post-treatment (see Section<br>12.2.1.1) | SAC |
| 16 | All Treated | AE8 | Listing of Adverse Events Leading to Withdrawal From Study | Add phase: Pre-treatment, on-<br>treatment, post-treatment (see Section<br>12.2.1.1) | SAC |
| 17 | All Treated | AE8 | Listing of Adverse Events Reported on the Day of Dosing | | SAC |
| Serious | Adverse Even | ts | | | |
| 18 | All Treated | AE8 | Listing of Fatal Serious Adverse Events | Add phase: Pre-treatment, on-<br>treatment, post-treatment (see Section<br>12.2.1.1) | SAC |
| 19 | All Treated | AE8 | Listing of Non-Fatal Serious Adverse Events | Add phase: Pre-treatment, on-<br>treatment, post-treatment (see Section<br>12.2.1.1) | SAC |
| 20 | All Treated | AE14 | Listing of Reasons for Considering as a Serious Adverse Event | | SAC |

| ICH and | ICH and Other Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Adverse Events of Special Interest | | | | | |
| 21 | All Treated | AE8 | Listing of Adverse Events Reported by the Investigator as Meeting the Criteria for Anaphylaxis | Add phase: Pre-treatment, on-treatment, post-treatment (see Section 12.2.1.1) Add injection reaction symptoms. | SAC |
| 22 | All Treated | AE8 | Listing of Adverse Events Defined by the Investigator as Systemic Reactions - Allergic (Type I Hypersensitivity) | Add phase: Pre-treatment, on-<br>treatment, post-treatment (see Section<br>12.2.1.1) Add injection reaction symptoms. | SAC |
| 23 | All Treated | AE8 | Listing of Adverse Events Defined by the Investigator as<br>Systemic Reactions – Other Systemic | Add phase: Pre-treatment, on-treatment, post-treatment (see Section 12.2.1.1) Add injection reaction symptoms. | SAC |
| 24 | All Treated | AE8 | Listing of Adverse Events Defined by the Investigator as Local Injection Site Reactions | Add phase: Pre-treatment, on-treatment, post-treatment (see Section 12.2.1.1) Add injection reaction symptoms. | SAC |
| 25 | All Treated | AE8 | Listing of Adverse Events Categorised as Serious Cardiac,<br>Vascular and Thromboembolic Events | Add phase: Pre-treatment, on-treatment, post-treatment (see Section 12.2.1.1) | SAC |
| 26 | All Treated | AE8 | Listing of Adverse Events Categorised as Serious Ischemic Events | Add phase: Pre-treatment, on-treatment, post-treatment (see Section 12.2.1.1) | SAC |

| ICH and | d Other Listings | <u> </u> | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 27 | All Treated | AE8 | Listing of Adverse Events Categorised as Malignancies | Add phase: Pre-treatment, on-<br>treatment, post-treatment (see Section<br>12.2.1.1) | SAC |
| 28 | All Treated | AE8 | Listing of Adverse Events Categorised as Opportunistic Infections | Add phase: Pre-treatment, on-<br>treatment, post-treatment (see Section<br>12.2.1.1) | SAC |
| Labora | tory | | | | |
| 29 | All Treated | LB5 | Listing of Haematology Data for Subjects with Abnormalities of Potential Clinical Concern | | SAC |
| 30 | All Treated | LB5 | Listing of Chemistry Data for Subjects with Abnormalities of Potential Clinical Concern | | SAC |
| Immun | ogenicity | | | | |
| 31 | All Treated | IMM2 | Listing of Immunogenicity Data for Subjects with at Least One Positive Screening Binding Assay | Include columns for Screening Binding<br>Assay, Confirmation Antibody Assay,<br>Confirmation Assay Titre,<br>Transient/Persistent, Neutralizing<br>Antibody Assay | SAC |
| User/De | evice Errors | <u>'</u> | | | |
| 32 | All Treated | LIST_ERR | Listing of User/Device Errors | List user/device errors for injections where full dose was not successfully administered only. | SAC |

### 12.11. Appendix 11: Example Mock Shells for Data Displays

Example TAB\_POP1
Protocol: MID204958


Population: All Subjects Enrolled

| Population | Liquid Autoinjector<br>(N=XX) | Liquid Safety Syringe (N=XX) | Lyophilised Vial (N=XX) | Total<br>(N=XXX) |
|---|---|---|---|---|
| All Subjects Enrolled | | | | XXX |
| Randomised | XXX | XXX | XXX | XXX |
| All Treated Subjects (Safety) | XXX (XX%) | XXX (XX%) | XXX (XX%) | XXX (XX%) |
| Pharmacokinetic | XXX (XX%) | XXX (XX%) | XXX (XX%) | XXX (XX%) |
| Pharmacodynamic | XXX (XX%) | XXX (XX%) | XXX (XX%) | XXX (XX%) |

204958


Example TAB\_POP2
Protocol: MID204958

Population: Randomised

| Population | Li | quid Autoing<br>(N=XX) | jector | Liq | uid Safety Syringe<br>(N=XX) | Ι | yophilised (N=XX) | Vial |
|---|---|---|---|---|---|---|---|---|
| _ | Arm | Abdomen | Thigh | Arm | Abdomen Thigh | Arm | Abdomen | Thigh |
| Randomised | XXX | XXX | XXX | XXX | xxx xxx | XXX | XXX | XXX |
| All Treated Subjects (Safety) | XXX (XX%) | XXX (XX%) | XXX (XX%) | XXX (XX% | ) XXX (XX%) XXX (XX%) | XXX (XX%) | XXX (XX%) | XXX (XX%) |
| Pharmacokinetic | XXX (XX%) | XXX (XX%) | XXX (XX%) | XXX (XX% | ) XXX (XX%) XXX (XX%) | XXX (XX%) | XXX (XX%) | XXX (XX%) |
| Pharmacodynamic | XXX (XX%) | XXX (XX%) | XXX (XX%) | XXX (XX% | ) XXX (XX%) XXX (XX%) | XXX (XX%) | XXX (XX%) | XXX (XX%) |

204958

Example TAB\_PK1

Protocol: MID204958 

Population: Pharmacokinetic

Table X.X Summary of Statistical Analysis of Derived Plasma Mepolizumab Pharmacokinetic Parameters

| Parameter | Test<br>treatment | Adjusted Geomet | tric Mean (SE (logs))<br>Reference [1] | Ratio<br>(Test/Ref) | 90% CI<br>for Ratio<br>(Test/Ref) |
|---|---|---|---|---|---|
| AUC(0-inf) (day*ug/mL) | Liquid Autoinjector | XX.XXX (X.XX) | XX.XXX (X.XX) | X.XXX | (X.XXX, X.XXX) |
| | Liquid Safety Syringe | XX.XXX (X.XX) | XX.XXX (X.XX) | X.XXX | (X.XXX, X.XXX) |
| AUC(0-t) (day*ug/mL) | Liquid Autoinjector | XX.XXX (X.XX) | XX.XXX (X.XX) | X.XXX | (X.XXX, X.XXX) |
| | Liquid Safety Syringe | XX.XXX (X.XX) | XX.XXX (X.XX) | X.XXX | (X.XXX, X.XXX) |
| Cmax (ug/mL) | Liquid Autoinjector | XX.XXX (X.XX) | XX.XXX (X.XX) | X.XXX | (X.XXX, X.XXX) |
| | Liquid Safety Syringe | XX.XXX (X.XX) | XX.XXX (X.XX) | X.XXX | (X.XXX, X.XXX) |

<sup>[1]</sup> Reference treatment = Lyophilised Vial.

Note: The estimates of the geometric mean are adjusted for injection site (arm, abdomen, thigh) and baseline weight (loge scale).

204958

Example TAB\_S1

Population: All Treated (Safety)

Table X.X

Summary Profile of On-Treatment Adverse Events Defined by the Investigator as Allergic (Type I Hypersensitivity) Reactions

| | | Liquid<br>Autoinjector<br>(N=XX) | Liquid Safety<br>Syringe<br>(N=XX) | Lyophilised<br>Vial<br>(N=XX) | Liquid<br>Total<br>(N=xx) | Total<br>(N=xx) |
|---|---|---|---|---|---|---|
| 1 | All Events | | | | | |
| | >= 1 event [1] | xx/xx (x%) | xx/xx (x%) | xx/xx (x%) | xx/xx (x%) | xx/xx (x%) |
| | 1 event | xx (x%) | xx (x%) | xx (x%) | xx (x%) | xx (x%) |
| | 2 events | xx (x%) | xx (x%) | xx (x%) | xx (x%) | xx (x%) |
| | 3 events | xx (x%) | xx (x%) | xx (x%) | xx (x%) | xx (x%) |
| | >=4 events | xx (x%) | xx (x%) | xx (x%) | xx (x%) | xx (x%) |
| 2 | Serious Events<br>>= 1 event [1] | xx/xx (x%) | xx/xx (x%) | xx/xx (x%) | xx/xx (x%) | xx/xx (x%) |
| 3 | <pre>Events considered related to investigational product &gt;= 1 event [1]</pre> | xx/xx (x%) | xx/xx (x%) | xx/xx (x%) | xx/xx (x%) | xx/xx (x%) |
| 4 | Intensity [1] | | | | | |
| | Mild | xx/xx (x%) | xx/xx (x%) | xx/xx (x%) | xx/xx (x%) | xx/xx (x%) |
| | Moderate | xx/xx (x%) | xx/xx (x%) | xx/xx (x%) | xx/xx (x%) | xx/xx (x%) |
| | Severe | xx/xx (x%) | xx/xx (x%) | xx/xx (x%) | xx/xx (x%) | xx/xx (x%) |
| 5 | Outcome [1] | | | | | |
| | Recovered/Resolving | xx/xx (x%) | xx/xx (x%) | xx/xx (x%) | xx/xx (x%) | xx/xx (x%) |
| | Recovering/Resolving | xx/xx (x%) | xx/xx (x%) | xx/xx (x%) | xx/xx (x%) | xx/xx (x%) |
| | Not recovered/Not Resolved | xx/xx (x%) | xx/xx (x%) | xx/xx (x%) | xx/xx (x%) | xx/xx (x%) |
| | Recovered/Resolved with sequelae | xx/xx (x%) | xx/xx (x%) | xx/xx (x%) | xx/xx (x%) | xx/xx (x%) |
| | Fatal | xx/xx (x%) | xx/xx (x%) | xx/xx (x%) | xx/xx (x%) | xx/xx (x%) |

<sup>[1]</sup> Information presented as number of events / number (%) subjects with at least one event. Subjects may be counted in more than one row.

<sup>[2]</sup> Cardiac History=Yes includes all subjects with any past medical condition under Cardiac Disorders

<sup>[3]</sup> Unable to categorise time since last dose as event time not reported

Example TAB\_S1 (Cont.)
Protocol: MID204958

Protocol: MID204958

Population: All Treated (Safety)

Table X.X

Summary Profile of On-Treatment Adverse Events Defined by the Investigator as Allergic (Type I Hypersensitivity) Reactions

| | | Liquid<br>Autoinjector<br>(N=XX) | Liquid Safety<br>Syringe<br>(N=XX) | Lyophilised<br>Vial<br>(N=XX) | Liquid<br>Total<br>(N=xx) | Total<br>(N=xx) |
|---|---|---|---|---|---|---|
| 6 | Action Taken [1] | | | | | _ |
| | Study treatment withdrawn | xx/xx (x%) | xx/xx (x%) | xx/xx (x%) | xx/xx (x%) | xx/xx (x%) |
| | Dose reduced | xx/xx (x%) | xx/xx (x%) | xx/xx (x%) | xx/xx (x%) | xx/xx (x%) |
| | Dose increased | xx/xx (x%) | xx/xx (x%) | xx/xx (x%) | xx/xx (x%) | xx/xx (x%) |
| | Dose not changed | xx/xx (x%) | xx/xx (x%) | xx/xx (x%) | xx/xx (x%) | xx/xx (x%) |
| | Dose interrupted/delayed | xx/xx (x%) | xx/xx (x%) | xx/xx (x%) | xx/xx (x%) | xx/xx (x%) |
| | Not applicable | xx/xx (x%) | xx/xx (x%) | xx/xx (x%) | xx/xx (x%) | xx/xx (x%) |
| 7 | Cardiac History [1][2] | | | | | |
| | Yes | xx/xx (x%) | xx/xx (x%) | xx/xx (x%) | xx/xx (x%) | xx/xx (x%) |
| | No | xx/xx (x%) | xx/xx (x%) | xx/xx (x%) | xx/xx (x%) | xx/xx (x%) |
| 8 | Anaphylaxis Criteria Met | | | | | |
| | Anaphylactic Criterion 1 | xx/xx (x%) | xx/xx (x%) | xx/xx (x%) | xx/xx (x%) | xx/xx (x%) |
| | Anaphylactic Criterion 2 | xx/xx (x%) | xx/xx (x%) | xx/xx (x%) | xx/xx (x%) | xx/xx (x%) |
| | Anaphylactic Criterion 3 | xx/xx (x%) | xx/xx (x%) | xx/xx (x%) | xx/xx (x%) | xx/xx (x%) |
| 9 | No. doses prior to event [1] | | | | | |
| | 1 | xx/xx (x%) | xx/xx (x%) | xx/xx (x%) | xx/xx (x%) | xx/xx (x%) |
| | 2 | xx/xx (x%) | xx/xx (x%) | xx/xx (x%) | xx/xx (x%) | xx/xx (x%) |
| | 3 | xx/xx (x%) | xx/xx (x%) | xx/xx (x%) | xx/xx (x%) | xx/xx (x%) |
| | etc. | | | | | |
| 10 | No. doses prior to first event | | | | | |
| | 1 | xx (x%) | xx (x%) | xx (x%) | xx (x%) | xx (x%) |
| | 2 | xx (x%) | xx (x%) | xx (x%) | xx (x%) | xx (x%) |
| | 3 | xx (x%) | xx (x%) | xx (x%) | xx (x%) | xx (x%) |
| | etc. | | | | | |

<sup>[1]</sup> Information presented as number of events / number (%) subjects with at least one event. Subjects may be counted in more than one row.

<sup>[2]</sup> Cardiac History=Yes includes all subjects with any past medical condition under Cardiac Disorders

 $<sup>\[3\]</sup>$  Unable to categorise time since last dose as event time not reported

Example TAB\_S1 (Cont.)
Protocol: MID204958


Population: All Treated (Safety)

Table X.X
Summary Profile of On-Treatment Adverse Events Defined by the Investigator as Allergic (Type I Hypersensitivity) Reactions

| | | Liquid<br>Autoinjector<br>(N=XX) | Liquid Safety<br>Syringe<br>(N=XX) | Lyophilised<br>Vial<br>(N=XX) | Liquid<br>Total<br>(N=xx) | Total<br>(N=xx) |
|---|---|---|---|---|---|---|
| 11 | Time since last dose to event | | | | | |
| | onset [1] | xx/xx (x%) | xx/xx (x%) | xx/xx (x%) | xx/xx (x%) | xx/xx (x%) |
| | <=1 hr | xx/xx (x%) | xx/xx (x%) | xx/xx (x%) | xx/xx (x%) | xx/xx (x%) |
| | 1-<6 hrs | xx/xx (x%) | xx/xx (x%) | xx/xx (x%) | xx/xx (x%) | xx/xx (x%) |
| | 6-<24 hrs | xx/xx (x%) | xx/xx (x%) | xx/xx (x%) | xx/xx (x%) | xx/xx (x%) |
| | >=24 hrs | xx/xx (x%) | xx/xx (x%) | xx/xx (x%) | xx/xx (x%) | xx/xx (x%) |
| | Missing[y] | | | | | |
| 12 | Time since last dose to first | | | | | |
| | event onset | xx (x%) | xx (x%) | xx (x%) | xx (x%) | xx (x%) |
| | <=1 hr | xx (x%) | xx (x%) | xx (x%) | xx (x%) | xx (x%) |
| | 1-<6 hrs | xx (x%) | xx (x%) | xx (x%) | xx (x%) | xx (x%) |
| | 6-<24 hrs | xx (x%) | xx (x%) | xx (x%) | xx (x%) | xx (x%) |
| | >=24 hrs | xx (x%) | xx (x%) | xx (x%) | xx (x%) | xx (x%) |
| | Missing [3] | | | | | |
| 13 | No. symptoms associated with event | | | | | |
| | [1] | xx/xx (x%) | xx/xx (x%) | xx/xx (x%) | xx/xx (x%) | xx/xx (x%) |
| | 0 symptoms | xx/xx (x%) | xx/xx (x%) | xx/xx (x%) | xx/xx (x%) | xx/xx (x%) |
| | 1 symptom | xx/xx (x%) | xx/xx (x%) | xx/xx (x%) | xx/xx (x%) | xx/xx (x%) |
| | 2-5 symptoms | xx/xx (x%) | xx/xx (x%) | xx/xx (x%) | xx/xx (x%) | xx/xx (x%) |
| | >5 symptoms | | | | | |
| 14 | Symptoms [1] | | | | | |
| | ABDOMINAL | xx/xx (x%) | xx/xx (x%) | xx/xx (x%) | xx/xx (x%) | xx/xx (x%) |
| | ANGIOEDEMA | xx/xx (x%) | xx/xx (x%) | xx/xx (x%) | xx/xx (x%) | xx/xx (x%) |
| | ARTHRALGIA | xx/xx (x%) | xx/xx (x%) | xx/xx (x%) | xx/xx (x%) | xx/xx (x%) |
| | etc | | | | | |

<sup>[1]</sup> Information presented as number of events / number (%) subjects with at least one event. Subjects may be counted in more than one row.

<sup>[2]</sup> Cardiac History=Yes includes all subjects with any past medical condition under Cardiac Disorders

<sup>[3]</sup> Unable to categorise time since last dose as event time not reported

204958

#### Programming Notes: -

Remove footnotes that are not relevant for the table.

Sections 1 - 6, 9, 10: Create for all adverse events of special interest

Sections 9 and 10: For studies longer than 1 year can consider the following categories: 1, 2, 3, 4, 5, 6, 7-12, 13-18,

19-24, >24

Section 7: Only for the following adverse events of special interest

Serious Cardiac, Vascular and Thromboembolic Events

Serious Ischemic Events

Section 8: Only for the following adverse events of special interest

Anaphylaxis

Systemic - Allergic (Type I Hypersensitivity)

Sections 11 - 14: Only for the following adverse events of special interest

Anaphylaxis

Systemic - Allergic (Type I Hypersensitivity) and Other Systemic

Systemic - Allergic (Type I Hypersensitivity)

Systemic - Other Systemic Local Injection Site Reactions

204958

Example TAB\_S2


Population: All Treated (Safety)

Table X
Summary of Binding Antibody Results by Visit

| Visit | Assay<br>Result | Liquid<br>Autoinjector<br>(N=XX) | Liquid Safety<br>Syringe<br>(N=XX) | Lyophilised<br>Vial<br>(N=XX) | Liquid<br>Total<br>(N=xx) | Total<br>(N=xx) |
|---|---|---|---|---|---|---|
| Screening | n | X | X | X | X | X |
| | NEGATIVE | X (XX%) | X (XX%) | X (XX%) | X (XX%) | X (XX%) |
| | POSITIVE | X (XX%) | X (XX%) | X (XX%) | X (XX%) | X (XX%) |
| Day 1 | n | X | X | X | X | X |
| | NEGATIVE | X (XX%) | X (XX%) | X (XX%) | X (XX%) | X (XX%) |
| | POSITIVE | X (XX%) | X (XX%) | X (XX%) | X (XX%) | X (XX%) |
| Day 29 | n | X | X | X | X | X |
| | NEGATIVE | X (XX%) | X (XX%) | X (XX%) | X (XX%) | X (XX%) |
| | POSITIVE | X (XX%) | X (XX%) | X (XX%) | X (XX%) | X (XX%) |
| | TRANSIENT POSITIVE | X (XX%) | X (XX%) | X (XX%) | X (XX%) | X (XX%) |
| | PERSISTENT POSITIVE | X (XX%) | X (XX%) | X (XX%) | X (XX%) | X (XX%) |

<sup>[1]</sup> A subject is considered positive if they have at least one positive post-baseline ADA result.

<sup>[2]</sup> Highest post-baseline titre.

204958

Example TAB\_S2 (Cont.)
Protocol: MID204958

Population: All Treated (Safety)

Table X
Summary of Binding Antibody Results by Visit

| Visit | Assay<br>Result | | Liquid<br>Autoinjector<br>(N=XX) | Liquid Safety<br>Syringe<br>(N=XX) | Lyophilised<br>Vial<br>(N=XX) | Liquid<br>Total<br>(N=xx) | Total (N=xx) |
|---|---|---|---|---|---|---|---|
| Day 43 | n | | X | X | Х | X | X |
| | NEGATIVE | | X (XX%) | X (XX%) | X (XX%) | X (XX%) | X (XX%) |
| | POSITIVE | | X (XX%) | X (XX%) | X (XX%) | X (XX%) | X (XX%) |
| | TRANSIENT POSITIVE | | X (XX%) | X (XX%) | X (XX%) | X (XX%) | X (XX%) |
| | PERSISTENT POSITIVE | | X (XX%) | X (XX%) | X (XX%) | X (XX%) | X (XX%) |
| Day 85 | n | | X | X | X | X | X |
| _ | NEGATIVE | | X (XX%) | X (XX%) | X (XX%) | X (XX%) | X (XX%) |
| | PERSISTENT POSITIVE | | X (XX%) | X (XX%) | X (XX%) | X (XX%) | X (XX%) |
| Any Post-<br>Baseline | n | | X | X | X | X | X |
| | NEGATIVE | | X (XX%) | X (XX%) | X (XX%) | X (XX%) | X (XX%) |
| | POSITIVE [1]<br>TRANSIENT POSITIVE<br>PERSISTENT POSITIVE | | X (XX%)<br>X (XX%)<br>X (XX%) | X (XX%)<br>X (XX%)<br>X (XX%) | X (XX%)<br>X (XX%)<br>X (XX%) | X (XX%)<br>X (XX%)<br>X (XX%) | X (XX%)<br>X (XX%)<br>X (XX%) |
| | Titre value [2] | Min.<br>Median<br>Max. | X<br>X.X<br>X | X<br>X.X<br>X | X<br>X.X<br>X | X<br>X.X<br>X | X<br>X.X<br>X |

<sup>[1]</sup> A subject is considered positive if they have at least one positive post-baseline ADA result.

<sup>[2]</sup> Highest post-baseline titre.

Example TAB\_S3

Protocol: MID204958 

Population: All Treated (Safety)

Table X
Summary of Neutralising Antibody Results by Visit

| Visit | Assay<br>Result | Liquid<br>Autoinjector<br>(N=XX) | Liquid Safety<br>Syringe<br>(N=XX) | Lyophilised<br>Vial<br>(N=XX) | Liquid<br>Total<br>(N=xx) | Total<br>(N=xx) |
|---|---|---|---|---|---|---|
| Caroonina | ~ | X | X | X | X | X |
| Screening | n<br>NEGATIVE | | | | | |
| | - | X (XX%) | X (XX%) | X (XX%) | X (XX%) | X (XX%) |
| | POSITIVE | X (XX%) | X (XX%) | X (XX%) | X (XX%) | X (XX%) |
| Day 1 | n | X | X | X | X | X |
| - 1 | NEGATIVE | X (XX%) | X (XX%) | X (XX%) | X (XX%) | X (XX%) |
| | POSITIVE | X (XX%) | X (XX%) | X (XX%) | X (XX%) | X (XX%) |
| D 0.0 | _ | 77 | 37 | 37 | 37 | 77 |
| Day 29 | n | X | X | X | X | X |
| | NEGATIVE | X (XX%) | X (XX%) | X (XX%) | X (XX%) | X (XX%) |
| | POSITIVE | X (XX%) | X (XX%) | X (XX%) | X (XX%) | X (XX%) |
| Day 43 | n | X | X | X | X | X |
| _ | NEGATIVE | X (XX%) | X (XX%) | X (XX%) | X (XX%) | X (XX%) |
| | POSITIVE | X (XX%) | X (XX%) | X (XX%) | X (XX%) | X (XX%) |
| Day 85 | n | X | X | X | X | X |
| Day 00 | NEGATIVE | X (XX%) | X (XX%) | X (XX%) | X (XX%) | X (XX%) |
| | POSITIVE | X (XX%) | X (XX%) | X (XX%) | X (XX%) | X (XX%) |
| | 10011110 | 21 (21210) | 21 (21210) | 21 (2121 0 ) | 21 (2121 0 ) | 21 (21210) |
| Any Post-Baseline | n | X | X | X | X | Χ |
| | NEGATIVE | X (XX%) | X (XX%) | X (XX%) | X (XX%) | X (XX%) |
| | POSITIVE [1] | X (XX%) | X (XX%) | X (XX%) | X (XX%) | X (XX%) |

<sup>[1]</sup> A subject is considered positive if they have at least one positive post-baseline neutralising antibody result.

204958

Example TAB\_PD1
Protocol: MID204958

Protocol: MID204958 
Population: Pharmacodynamic

| Treatment | N | Visit | n | Geom.<br>Mean | 95% CI<br>(Lower,Upper) | SD (logs) | Min. | Median | Max. |
|---|---|---|---|---|---|---|---|---|---|
| Treatment | 14 | VIDIC | 11 | ncan | (Hower, opper) | 5D (1095) | 11111. | Healan | nax. |
| Lyophilised Vial | XX | Day 1 | XX | xxxx.xx | (xxxx.xx,xxxx.xx) | xx.xxx | XX.X | xxxx.xx | xx.x |
| | | Day 3 | XX | XXXX.XX | (xxxx.xx, xxxx.xx) | XX.XXX | XX.X | XXXX.XX | XX.X |
| | | Day 5 | XX | XXXX.XX | (xxxx.xx,xxxx.xx) | XX.XXX | XX.X | XXXX.XX | XX.X |
| | | Day 10 | XX | XXXX.XX | (xxxx.xx, xxxx.xx) | XX.XXX | XX.X | XXXX.XX | XX.X |
| | | Day 29 | XX | XXXX.XX | (xxxx.xx, xxxx.xx) | XX.XXX | XX.X | XXXX.XX | XX.X |
| | | Day 57 | XX | XXXX.XX | (xxxx.xx, xxxx.xx) | XX.XXX | XX.X | XXXX.XX | XX.X |
| | | Day 85 | XX | XXXX.XX | (xxxx.xx,xxxx.xx) | XX.XXX | XX.X | XXXX.XX | XX.X |
| Liquid Autoinjector | XX | Day 1 | XX | xxxx.xx | (xxxx.xx,xxxx.xx) | xx.xxx | xx.x | xxxx.xx | XX.X |
| | | Day 3 | XX | XXXX.XX | (xxxx.xx,xxxx.xx) | XX.XXX | XX.X | XXXX.XX | XX.X |
| | | Day 5 | XX | XXXX.XX | (xxxx.xx,xxxx.xx) | XX.XXX | XX.X | XXXX.XX | XX.X |
| | | Day 10 | XX | XXXX.XX | (xxxx.xx,xxxx.xx) | XX.XXX | XX.X | XXXX.XX | XX.X |
| | | Day 29 | XX | XXXX.XX | (xxxx.xx,xxxx.xx) | XX.XXX | XX.X | XXXX.XX | XX.X |
| | | Day 57 | XX | XXXX.XX | (xxxx.xx, xxxx.xx) | XX.XXX | XX.X | XXXX.XX | XX.X |
| | | Day 85 | XX | xxxx.xx | (xxxx.xx,xxxx.xx) | XX.XXX | XX.X | XXXX.XX | XX.X |
| Liquid Safety Syringe | XX | Day 1 | XX | xxxx.xx | (xxxx.xx,xxxx.xx) | XX.XXX | xx.x | xxxx.xx | XX.X |
| | | Day 3 | XX | xxxx.xx | (xxxx.xx,xxxx.xx) | XX.XXX | XX.X | xxxx.xx | XX.X |
| | | Day 5 | XX | xxxx.xx | (xxxx.xx,xxxx.xx) | XX.XXX | XX.X | xxxx.xx | XX.X |
| | | Day 10 | XX | xxxx.xx | (xxxx.xx, xxxx.xx) | XX.XXX | XX.X | xxxx.xx | XX.X |
| | | Day 29 | XX | xxxx.xx | (xxxx.xx, xxxx.xx) | XX.XXX | XX.X | xxxx.xx | XX.X |
| | | Day 57 | XX | xxxx.xx | (xxxx.xx, xxxx.xx) | XX.XXX | XX.X | xxxx.xx | XX.X |
| | | Day 85 | XX | XXXX.XX | (xxxx.xx,xxxx.xx) | XX.XXX | XX.X | XXXX.XX | XX.X |

204958

Example TAB\_PD2 Protocol: MID204958

Protocol: MID204958 
Population: Pharmacodynamic

Table X
Summary of Ratio to Baseline Blood Eosinophils

| Treatment | N | Visit | n | Geom.<br>Mean | 95% CI<br>(Lower,Upper) | SD (logs) | Min. | Median | Max. |
|---|---|---|---|---|---|---|---|---|---|
| Lyophilised Vial | XX | Day 3 | XX | XXXX.XX | (xxxx.xx,xxxx.xx) | XX.XXX | XX.X | XXXX.XX | XX.X |
| | | Day 5 | XX | XXXX.XX | (xxxx.xx,xxxx.xx) | XX.XXX | XX.X | XXXX.XX | XX.X |
| | | Day 10 | XX | XXXX.XX | (xxxx.xx, xxxx.xx) | XX.XXX | XX.X | XXXX.XX | XX.X |
| | | Day 29 | XX | XXXX.XX | (xxxx.xx, xxxx.xx) | XX.XXX | XX.X | XXXX.XX | XX.X |
| | | Day 57 | XX | XXXX.XX | (xxxx.xx, xxxx.xx) | XX.XXX | XX.X | XXXX.XX | XX.X |
| | | Day 85 | XX | xxxx.xx | (xxxx.xx, xxxx.xx) | XX.XXX | XX.X | XXXX.XX | XX.X |
| Liquid Autoinjector | XX | Day 3 | XX | xxxx.xx | (xxxx.xx,xxxx.xx) | XX.XXX | XX.X | XXXX.XX | XX.X |
| 1 | | Day 5 | XX | xxxx.xx | (xxxx.xx, xxxx.xx) | XX.XXX | XX.X | xxxx.xx | XX.X |
| | | Day 10 | XX | xxxx.xx | (xxxx.xx, xxxx.xx) | XX.XXX | XX.X | xxxx.xx | XX.X |
| | | Day 29 | XX | xxxx.xx | (xxxx.xx,xxxx.xx) | xx.xxx | XX.X | xxxx.xx | XX.X |
| | | Day 57 | XX | xxxx.xx | (xxxx.xx,xxxx.xx) | xx.xxx | XX.X | xxxx.xx | XX.X |
| | | Day 85 | XX | xxxx.xx | (xxxx.xx,xxxx.xx) | xx.xx | XX.X | xxxx.xx | XX.X |
| Liquid Safety Syringe | XX | D211 3 | XX | XXXX.XX | (0000 00 0000 00) | xx.xxx | xx.x | VVVV VV | XX.X |
| Liquid Salety Syllinge | ΛΛ | Day 3 | | | (xxxx.xx, xxxx.xx) | | | XXXX.XX | |
| | | Day 5 | XX | XXXX.XX | (xxxx.xx, xxxx.xx) | XX.XXX | XX.X | XXXX.XX | XX.X |
| | | Day 10 | XX | XXXX.XX | (xxxx.xx, xxxx.xx) | XX.XXX | XX.X | XXXX.XX | XX.X |
| | | Day 29 | XX | XXXX.XX | (xxxx.xx,xxxx.xx) | XX.XXX | XX.X | XXXX.XX | XX.X |
| | | Day 57 | XX | XXXX.XX | (xxxx.xx,xxxx.xx) | XX.XXX | XX.X | XXXX.XX | XX.X |
| | | Day 85 | XX | XXXX.XX | (xxxx.xx, xxxx.xx) | XX.XXX | XX.X | XXXX.XX | XX.X |

204958

Example TAB\_PD3

Protocol: MID204958 

Population: Pharmacodynamic

Table X.X Summary of Statistical Analysis of Ratio to Baseline Blood Eosinophils

| Test<br>treatment | Visit | Adjusted Geome | tric Mean (SE (logs)) Reference [1] | Ratio<br>(Test/Ref) | 95% CI<br>for Ratio<br>(Test/Ref) |
|---|---|---|---|---|---|
| Liquid Autoinjector | Day 3<br>Day 5<br>Day 10<br>Day 29<br>Day 57 | XX.XXX (X.XX)<br>XX.XXX (X.XX)<br>XX.XXX (X.XX)<br>XX.XXX (X.XX)<br>XX.XXX (X.XX) | XX.XXX (X.XX)<br>XX.XXX (X.XX)<br>XX.XXX (X.XX)<br>XX.XXX (X.XX)<br>XX.XXX (X.XX) | X.XXX<br>X.XXX<br>X.XXX<br>X.XXX<br>X.XXX | (X.XXX, X.XXX)<br>(X.XXX, X.XXX)<br>(X.XXX, X.XXX)<br>(X.XXX, X.XXX)<br>(X.XXX, X.XXX) |
| Liquid Safety Syringe | Day 85 Day 3 Day 5 Day 10 Day 29 Day 57 Day 85 | XX.XXX (X.XX) XX.XXX (X.XX) XX.XXX (X.XX) XX.XXX (X.XX) XX.XXX (X.XX) XX.XXX (X.XX) XX.XXX (X.XX) | XX.XXX (X.XX) XX.XXX (X.XX) XX.XXX (X.XX) XX.XXX (X.XX) XX.XXX (X.XX) XX.XXX (X.XX) XX.XXX (X.XX) | X.XXX<br>X.XXX<br>X.XXX<br>X.XXX<br>X.XXX<br>X.XXX | (X.XXX, X.XXX) (X.XXX, X.XXX) (X.XXX, X.XXX) (X.XXX, X.XXX) (X.XXX, X.XXX) (X.XXX, X.XXX) (X.XXX, X.XXX) |

#### [1] Reference treatment = Lyophilised Vial.

Note: The estimates of the geometric mean are adjusted for baseline blood eosinophil count (loge scale), injection site (arm, abdomen, thigh) and baseline weight (loge scale).

204958

Example TAB\_AI

Protocol: MID204958 

Population: All Treated Subjects (Safety)

Table X.X

Summary of Injection Assessment - Liquid Autoinjector

| | | Liquid Autoinjector (N=XX) |
|---|---|---|
| Was the full dose successfully administered? | Yes<br>No | XX (XX%)<br>XX (XX%) |
| User Errors | Incorrect injection site Pen was not pushed all the way down and held Pen was pulled away before end of injection Evidence of liquid leaking from the injection site Other | XX (XX%) XX (XX%) XX (XX%) XX (XX%) XX (XX%) |
| Device Errors | Pen leaking Components broken/cracked Cannot push the needle guard down to activate Pen does not activate (after pressing the needle guard down) Delivery stops before the end of injection Other | XX (XX%) XX (XX%) XX (XX%) XX (XX%) XX (XX%) XX (XX%) |

Example TAB\_SS

Protocol: MID204958 

Population: All Treated Subjects (Safety)

Table X.X

Summary of Injection Assessment - Liquid Safety Syringe

| | Liquid | | ety Syringe<br>XX) |
|---|---|---|---|
| Was the full dose successfully administered? | Yes<br>No | | (XX%)<br>(XX%) |
| User Errors | Incorrect injection site Needle not full inserted into site Plunger not slowly pushed down Plunger not pushed all the way down until the stopper reaches bottom of syringe Thumb not moved up, plunger not risen and needle guard not activated Evidence of liquid leaking from injection site Other | XX<br>XX<br>XX | (XX%)<br>(XX%)<br>(XX%)<br>(XX%)<br>(XX%)<br>(XX%) |
| Device Errors | Syringe leaking<br>Components broken/cracked<br>Cannot push the plunger rod down<br>Other | XX<br>XX | (XX%)<br>(XX%)<br>(XX%) |

Example LIST\_ERR

Abdomen

Protocol: MID204958 

Population: All Treated Subjects (Safety)

Table X.X

Listing of User/Device Errors

| Treatment/<br>Injection Site | Site Id./<br>Unique<br>Subject Id. | Was the Full Dose<br>Successfully Administered? | User/Device Error |
|---|---|---|---|
| Liquid Autoinjector/<br>Arm | XXXXXX/<br>MID204958.XXXXXX | No | Delivery stops before end of injection |
| | XXXXXX/<br>MID204958.XXXXXX | No | Incorrect injection site selected - specify Pen leaking |
| Liquid Safety Syringe/ | XXXXXX/ | No | Incorrect injection site selected - specify |

userid: /arenv/arprod/compound/study/final/drivers/drivername.sas DDMMMYYYY HH:MM

MID204958.XXXXXX

Example FIG\_PK1

Protocol: MID204958 

Population: Pharmacokinetic

Figure X.X

Individual Subject (+Geometric Mean and 95% CI) Derived Plasma Mepolizumab PK Parameters by Treatment

Parameter: AUC (mcg\*days/mL)



Example FIG\_PK2

Protocol: MID204958 
Population: Pharmacokinetic

Figure X.X Individual Subject (+Geometric Mean and 95% CI) Derived Plasma Mepolizumab PK Parameters by Treatment and Injection Site

Parameter: AUC (mcg\*days/mL)



Example FIG\_PK3

Protocol: MID204958


Population: Pharmacokinetic

Figure X.X

Individual Subject (+Geometric Mean and 95% CI) Derived Plasma Mepolizumab PK Parameters by Baseline Body Weight Category and Treatment

Parameter: AUC (mcg\*days/mL)



Example FIG\_PK4

Protocol: MID204958 
Population: Pharmacokinetic

Figure X.X

Individual Subject (+Geometric Mean and 95% CI) Derived Plasma Mepolizumab PK Parameters by Baseline Body Weight Category, Treatment and Injection Site

Parameter: AUC (mcg\*days/mL), Baseline Body Weight: <70 kg



Example FIG\_PK5

Protocol: MID204958 

Population: Pharmacokinetic

Figure X.X

Adjusted Geometric Means and Treatment Ratios (90% CI) for Primary Analysis of Derived Plasma Mepolizumab PK Parameters

Parameter: AUC (mcg\*days/mL)



Example FIG\_PD1

Protocol: MID204958 

Population: All Treated (Safety)

Figure X.X Summary of Adjusted Geometric Mean (95% CI) Ratio to Baseline Blood Eosinophils by Visit



Example FIG\_PD2

Protocol: MID204958 

Population: All Treated (Safety)  $\mbox{ Figure X.X}$ 

Summary of Adjusted Treatment Ratios (95% CI) for Ratio to Baseline Blood Eosinophils by Visit

